

#### CLINICAL STUDY PROTOCOL

Study Title: A Multicenter, Randomized, Phase 3, Open-Label Study to

Investigate the Efficacy and Safety of Sofosbuvir/Velpatasvir ± Ribavirin for 12 Weeks in Subjects with Chronic HCV Infection and

**Decompensated Cirrhosis** 

Sponsor: Gilead Sciences, Inc.

333 Lakeside Drive

Not Applicable

Foster City, CA 94404, USA

IND Number: This is a non-IND study

EudraCT Number:

Clinical Trials.gov

Identifier: Not Available

Indication: Hepatitis C Virus Infection

Protocol ID: GS-US-342-4019

Gilead Study Director Name:

Telephone: PPD Fax: PPD

Email: PPU

Gilead Medical Name: Anu Osinusi, MD, MPH

Monitor: Telephone: PPD Fax: PPD

Email:

Protocol Version/Date: Original: 03 October 2016

Amendment 1: 17 November 2016

PPD

# CONFIDENTIALITY STATEMENT

The information contained in this document, particularly unpublished data, is the property or under control of Gilead Sciences, Inc., and is provided to you in confidence as an investigator, potential investigator, or consultant, for review by you, your staff, and an applicable Institutional Review Board or Independent Ethics Committee. The information is only to be used by you in connection with authorized clinical studies of the investigational drug described in the protocol. You will not disclose any of the information to others without written authorization from Gilead Sciences, Inc., except to the extent necessary to obtain informed consent from those persons to whom the drug may be administered.

# TABLE OF CONTENTS

| LIST O | F IN-TEXT T | TABLES | 5 |
|---|---|---|---|
| PROTO | OCOL SYNOI | PSIS | 6 |
| GLOSS | SARY OF AB | BREVIATIONS AND DEFINITION OF TERMS | 11 |
| 1. IN | INTRODUCTION | | 16 |
| 1. | 1. Backgro | 1. Background | |
| | 1.1.1. HCV Infection in Japan | | 16 |
| 1. | 2. Sofosbu | nvir/Velpatasvir Fixed-Dose Combination | 17 |
| 1. | 3. Informa | ation about Ribavirin | 17 |
| 1. | 4. Rationa | ile for This Study | 17 |
| 1. | <ol><li>Rationa</li></ol> | le for Dose Selection of SOF/VEL | 18 |
| 1. | | | |
| 1. | 7. Risk/Be | Risk/Benefit Assessment for the Study | |
| 1. | 8. Complia | ance | 19 |
| 2. O | BJECTIVES. | | 20 |
| 3. ST | TUDY DESIG | GN | 21 |
| 3. | 1. Study E | Design | 21 |
| 3. | 12/40 CHARLES THE STREET | Freatments | |
| 3. | The state of the s | n of Treatment | |
| 3. | | g Rules and Discontinuation Criteria | |
| | 3.4.1. | Toxicity-Based Stopping Criteria | |
| | 3.4.2. | Virologic Response-Based Treatment Stopping Criteria | |
| 3. | | | 23 |
| 3. | 6. PPD | | 24 |
| 4. SI | UBJECT POP | ULATION | 26 |
| 4. | 1. Number | 26 | |
| 4. | | Inclusion Criteria. | |
| 4. | 3. Exclusion | 27 | |
| 5. IN | VESTIGATI | ONAL MEDICINAL PRODUCTS | 30 |
| 5. | 1. Randon | nization, Blinding and Treatment Codes | 30 |
| 5. | 2. Descrip | otion and Handling of SOF/VEL FDC | 30 |
| | 5.2.1. | Formulation | 30 |
| | 5.2.2. | SOF/VEL FDC Packaging and Labeling | 30 |
| | 5.2.3. | SOF/VEL FDC Storage and Handling | 31 |
| | 5.2.4. | Dosage and Administration of SOF/VEL FDC | |
| 5. | <ol><li>Descrip</li></ol> | otion and Handling of Ribavirin (RBV) | 31 |
| | 5.3.1. | Formulation | |
| | 5.3.2. | RBV Packaging and Labeling | |
| | 5.3.3. | RBV Storage and Handling | |
| | 5.3.4. | Dosage and Administration of RBV) | |
| 5. | | | |
| | 5.5. Study Drug Adherence and Drug Accountability | | |
| 250 | | | |
| 5. | .7. Accountability for Study Drug | | |
| | 5.7.1. | Study Drug Return or Disposal | 35 |
| 6. ST | TUDY PROC | EDURES | 36 |

| | 6.1. | Screening Visit | 36 |
|---|---|---|---|
| | | 6.1.1. Day 1 Assessments | 38 |
| | 6.2. | Study Drug Administration | 39 |
| | 6.3. | Close Monitoring During Early Phase of Treatment for Subjects with CPT C Cirrhosis | 39 |
| | 6.4. | Treatment Assessments (± 3 days) | 39 |
| | | 6.4.1. Weeks 1, 3, 5, 6, 7, 9, 10, and 11 (± 3 days) | |
| | | 6.4.2. Week 2 (± 3 days) | 40 |
| | | 6.4.3. Weeks 4 and 8 (± 3 days) | |
| | | 6.4.4. Week 12 (± 3 days) | |
| | 6.5. | Posttreatment Assessments (± 5 days) | |
| | | 6.5.1. Posttreatment Week 4 (± 5 days) | |
| | | 6.5.2. Posttreatment Week 12 (± 5 days) | |
| | | 6.5.3. Posttreatment Week 24 (± 5 days) | |
| | 6.6. | Early Termination (ET) | |
| | 6.7. | Unscheduled Visit | |
| | 6.8. | Procedures and Specifications. | |
| | 0.0. | 6.8.1. Clinical Laboratory Analytes | |
| | | 6.8.2. Medical History | |
| | | 6.8.3. Complete Physical Examination. | |
| | | 6.8.4. Vital Signs | |
| | | 6.8.5. 12-Lead ECG. | |
| | | 6.8.6. Health Related Quality of Life (HRQoL) | |
| | | 6.8.7. MELD and CPT Score Calculations | |
| | | 6.8.8. Creatinine Clearance | |
| | | 6.8.9. Viral RNA Sequencing / Phenotyping Sample | |
| | | 6.8.10. HBV DNA Sample | |
| | | 6.8.11. Single Pharmacokinetic (PK) Sample | |
| | | 6.8.12. Pregnancy Testing | |
| | | 6.8.13. IL28B Testing | |
| | | • | |
| | 6.0 | 6.8.15. Genomic Testing | |
| | 6.9. | End of Study. | |
| | 6.10. | Post Study Care | 31 |
| 7. | ADV | ERSE EVENTS AND TOXICITY MANAGEMENT | 52 |
| | 7.1. | Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events | 52 |
| | 7.1. | 7.1.1. Adverse Events | |
| | | 7.1.2. Serious Adverse Events | |
| | | 7.1.2. Serious Adverse Events | |
| | | Adverse Events or Serious Adverse Events | |
| | 7.2 | Assessment of Adverse Events and Serious Adverse Events | |
| | 7.2. | | |
| | | 7.2.1. Assessment of Causality for Study Drugs and Procedures | |
| | 7.2 | 7.2.2. Assessment of Severity | 34 |
| | 7.3. | Investigator Requirements and Instructions for Reporting Adverse Events and Serious | <i>-</i> 1 |
| | 7.4 | Adverse Events to Gilead or CRO | |
| | 7.4. | Gilead Reporting Requirements | |
| | 7.5. | Toxicity Management | |
| | 7.6 | 7.5.1. RBV Dose Adjustments | |
| | 7.6. | Special Situations Reports | |
| | | 7.6.1. Definitions of Special Situations | |
| | | 7.6.2. Instructions for Reporting Special Situations | 58 |
| 8. | STAT | ISTICAL CONSIDERATIONS | 60 |
| | 8.1. | Analysis Objectives and Endpoints | 60 |
| | 0.1. | Thingsis Cojectives and Diaponies | 00 |

| | | 8.1.1. | Analysis Objectives | |
|---|---|---|---|---|
| | | 8.1.2. | Primary Endpoint | |
| | | 8.1.3. | Secondary Endpoint | 61 |
| | | 8.1.4. | Other Endpoints of Interest | 61 |
| | 8.2. | Analys | s Conventions. | 61 |
| | | 8.2.1. | Analysis Sets | 61 |
| | 8.3. | | andling Conventions | |
| | 8.4. | Demog | raphic Data and Baseline Characteristics | 63 |
| | 8.5. | Efficac | y Analysis | 63 |
| | | 8.5.1. | Primary Analysis | 63 |
| | | 8.5.2. | Secondary Analyses | 63 |
| | 8.6. | Safety A | Analysis | 64 |
| | | 8.6.1. | Extent of Exposure | 64 |
| | | 8.6.2. | Adverse Events | 64 |
| | | 8.6.3. | Laboratory Evaluations | 65 |
| | | 8.6.4. | Other Safety Evaluations | 65 |
| | 8.7. | Pharma | cokinetic Analysis | 65 |
| | 8.8. | | Size | |
| | 8.9. | Data M | onitoring Committee | 66 |
| 9. | RESE | ONSIBIL | ITIES | 67 |
| | 9.1. | Investig | gator Responsibilities | 67 |
| | | 9.1.1. | Good Clinical Practice | 67 |
| | | 9.1.2. | Institutional Review Board (IRB)/Independent Ethics Committee (IEC) | |
| | | | Review and Approval | 67 |
| | | 9.1.3. | Informed Consent | 67 |
| | | 9.1.4. | Confidentiality | 68 |
| | | 9.1.5. | Study Files and Retention of Records | 68 |
| | | 9.1.6. | Case Report Forms | 69 |
| | | 9.1.7. | Study Drug Accountability and Return | 70 |
| | | 9.1.8. | Inspections | 70 |
| | | 9.1.9. | Protocol Compliance | 70 |
| | 9.2. | Sponso | r Responsibilities | 71 |
| | | 9.2.1. | Protocol Modifications | 71 |
| | | 9.2.2. | Study Report and Publications | 71 |
| | 9.3. | Joint In | vestigator/Sponsor Responsibilities | |
| | | 9.3.1. | Access to Information for Monitoring | |
| | | 9.3.2. | Access to Information for Auditing or Inspections | |
| | | 9.3.3. | Study Discontinuation | 72 |
| 10. | REFE | ERENCES | | 73 |
| 11. | APPE | ENDICES | | 76 |
| | Anne | ndiv 1 | Investigator Signature Page | 77 |
| | Appendix 1. Appendix 2. | | Study Procedures Table | |
| | | | GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities | |
| | | | Pregnancy Precautions, Definition for Female of Childbearing Potential, and | 01 |
| | | | Contraceptive Requirements | 103 |

# LIST OF IN-TEXT TABLES

| Table 5-1. | Dosing and Administration of RBV | 32 |
|---|---|---|
| Table 5-2. | Disallowed and Concomitant Medications to be Used with Caution | |
| Table 6-1. | Child-Pugh-Turcotte Classification of the severity of cirrhosis | 48 |
| Table 7-1 | RBV Dose Reduction Recommendations | |

# PROTOCOL SYNOPSIS

# Gilead Sciences, Inc. 333 Lakeside Drive Foster City, CA 94404, USA

| Study Title: IND Number: | A Multicenter, Randomized, Phase 3, Open-Label Study to Investigate the Efficacy and Safety of Sofosbuvir/Velpatasvir ± Ribavirin for 12 Weeks in Subjects with Chronic HCV Infection and Decompensated Cirrhosis This is a non-IND study |
|---|---|
| EudraCT Number:<br>Clinical Trials.gov<br>Identifier: | Not Available Not Available |
| Study Centers Planned: | Approximately 30 centers in Japan |

# **Objectives:**

The primary objectives of this study are:

- To evaluate the antiviral efficacy of therapy with sofosbuvir/velpatasvir (SOF/VEL) fixed-dose combination (FDC) with or without ribavirin for 12 weeks as measured by the proportion of subjects with sustained virologic response 12 weeks after cessation of treatment (SVR12)
- To evaluate the safety and tolerability of each treatment regimen

The secondary objectives of this study are:

- To determine the proportion of subjects who attain SVR at 4 and 24 weeks after cessation of treatment (SVR4 and SVR24)
- To evaluate the proportion of subjects with virologic failure
- To evaluate therapeutic efficacy as measured by the change of CPT score and MELD score
- To evaluate the kinetics of circulating HCV RNA during treatment and after cessation of treatment
- To evaluate the emergence of viral resistance to SOF and VEL during treatment and after cessation of treatment

The exploratory objectives of this study are:



# Study Design:

This is a multicenter, randomized, open-label study in subjects with chronic HCV infection with decompensated cirrhosis.

Approximately 100 subjects will be randomized (1:1) to one of the following two treatment groups:

- SOF/VEL (400/100 mg) for 12 weeks (n=50)
- SOF/VEL (400/100 mg) with RBV for 12 weeks (n=50)

Randomization will be stratified by Child-Pugh-Turcotte (CPT) class at Screening (CPT B/ CPT C) and HCV genotype (genotype 1/ non-genotype 1). For the purposes of randomization, a subject with non-definitive or mixed HCV genotype results by central laboratory analysis will be considered non-genotype 1. At least 15 subjects will have non-genotype 1 HCV infection. Approximately 10% of subjects will have CPT C (score 10-12) cirrhosis.

Initially only subjects with CPT B cirrhosis (score 7-9) at Screening will be enrolled. Enrollment of subjects with CPT C cirrhosis at Screening (score 10-12) will begin after the Data Monitoring Committee (DMC) has reviewed accumulated safety data from the first 20 subjects through 4 weeks of treatment (or early treatment discontinuation) and concluded that these data support enrollment of subjects with CPT C cirrhosis.

Number of Subjects Planned: Approximately 100 subjects

Target Population:

Adults with chronic HCV infection and decompensated cirrhosis.

Duration of Treatment:

Subjects will be treated for 12 weeks.

Diagnosis and Main Eligibility Criteria: Chronic HCV infected male and non-pregnant/non-lactating female subjects aged 20 years or older with decompensated cirrhosis.

Study Procedures/ Frequency: All subjects will complete the following study visits: Screening, Day 1, on-treatment visits at the end of Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12, and posttreatment visits at Weeks 4, 12, and 24 after completion of treatment.

Screening assessments will be completed within 28 days of the Day 1 visit. The screening window can be extended up to 42 days for subjects for extenuating circumstances with sponsor approval.

Screening assessments will include obtaining informed consent, physical examination, medical history, height, weight, vital signs, 12-lead electrocardiogram (ECG), adverse events (AEs) related to screening procedures, concomitant medications, laboratory tests (including hematology, chemistry, and coagulation), calculation of CPT and Model for End Stage Liver Disease (MELD) scores, HCV RNA, HCV genotyping, serology (HIV, HCV, HBV), Fibrotest<sup>®</sup>, liver imaging to exclude hepatocellular carcinoma (HCC) (if appropriate historical results are not available), serum β-hCG (females of child bearing potential only), and urinalysis.

Single 12-lead ECGs will be collected at Screening and Day 1 (prior to study drug administration).

On-treatment assessments include physical examination, weight, vital signs, AEs, concomitant medications, review of study drugs adherence and drug accountability, safety laboratory tests (including hematology, chemistry, coagulation), calculation of CPT and MELD scores, HCV RNA, IL28B genotyping, pharmacokinetic samples, health-related quality of life (HRQoL) surveys, and urine pregnancy tests (females of child bearing potential only). Subjects with CPT C cirrhosis at Screening will undergo close monitoring in the early phase of treatment.

Posttreatment assessments include physical examination, weight, vital signs, AEs and concomitant medications, safety laboratory tests (including hematology, chemistry, coagulation), calculation of CPT and MELD scores, HCV RNA, HRQoL surveys, and urine pregnancy tests (females of childbearing potential only).

HRQoL surveys (SF-36, CLDQ-HCV, FACIT-F, and WPAI) will be conducted at Day 1, on-treatment Week 12 or Early Termination (ET; if applicable), and posttreatment Week 12.

Samples for HCV RNA sequencing / phenotyping and HBV DNA will be collected at Day 1 (except HBV DNA) and on-treatment Weeks 2, 4, 8, and 12 or ET and post-treatment Weeks 4, 12, and 24. Samples will be collected during on-treatment Weeks 2, 4, 8, and 12 or ET for pharmacokinetic (PK) analysis of study drugs.

PPD .

# Test Product, Dose, and Mode of Administration:

SOF/VEL fixed dose combination (FDC) is manufactured as a 400/100 mg tablet for oral administration. Subjects will take 1 tablet daily with or without food.

Ribavirin (REBETOL<sup>®</sup>, RBV) is manufactured as a 200 mg capsule. Subjects with CPT B cirrhosis at Screening will take weight-based RBV every day (600-1000 mg/day in a divided daily dose). Subjects with CPT C cirrhosis at Screening will take 600 mg/day in a divided daily dose. The subject will take the morning dose of RBV with the SOF/VEL tablet and with food. The evening dose of RBV will be taken alone with food.

# Reference Therapy, Dose, and Mode of Administration:

None

# Criteria for Evaluation:

Safety: AEs and laboratory tests will be collected throughout the study.

Efficacy: Efficacy will be evaluated using scheduled assessments of HCV RNA

performed using COBAS® AmpliPrep®/COBAS® TaqMan® HCV

Quantitative Test, v2.0.

Efficacy will also be evaluated using scheduled assessments of CPT

and MELD scores.

Pharmacokinetics: A single PK blood sample will be collected at each on-treatment visit

for all subjects. The PK of SOF (and metabolites), VEL and RBV

may be assessed.

#### **Statistical Methods:**

The primary efficacy endpoint for the study is SVR12 in all randomized and treated subjects.

In the primary efficacy analysis, the SVR12 rate for subjects in each of the two treatment groups will be compared to the spontaneous clearance rate of 1% using the two-sided exact one-sample binomial test with Bonferroni alpha adjustment (each at significance level of 0.025).

Secondary endpoints include SVR4 and SVR24; proportion of subjects who have HCV RNA < LLOQ by visit while on study treatment; absolute and change from baseline in HCV RNA through end of treatment; virologic failure; and change from baseline in MELD and CPT scores.


A sample size of 50 subjects in each treatment group will provide over 99% power to detect at least 40% improvement in SVR12 rate from the assumed spontaneous rate of 1% or less using a two-sided exact one-sample binomial test at significance level of 0.025.

This study will be conducted in accordance with ICH Good Clinical Practice (GCP), and J-GCP (Ministerial Ordinance on Good Clinical Practice for Drugs), and all applicable regulatory requirements, including archiving of essential documents.

# GLOSSARY OF ABBREVIATIONS AND DEFINITION OF TERMS

° C degrees Celsius ° F degrees Fahrenheit

Ab antibody

ABW actual body weight
ADD Attention deficit disorder

AE(s) adverse event(s)

ALT alanine aminotransferase (also SGPT)

ANC absolute neutrophil count

aPTT activated partial thromboplastin time
AST aspartate aminotransferase (also SGOT)

ASV asunaprevir

AUC area under the curve AV atrioventricular

BLQ below limit of quantification

BMD bone mineral density
BMI body mass index
BW body weight

CD4+ cluster of differentiation 4+
CFR Code of Federal Regulations
CHF congestive heart failure
CI confidence interval
CICr creatinine clearance

CLDQ-HCV Chronic Liver Disease Questionnaire

cm<sup>2</sup> square centimeter

Cmax the maximum observed serum/plasma/peripheral blood mononuclear (PBMC)

concentration of drug

CNS Central nervous system
CPT Child-Pugh-Turcotte

CRO contract (or clinical) research organization

CSR clinical study report

CVA Cerebral vascular accident
DAA direct-acting antiviral

DCV daclatasvir dL Deciliter

DMC Data Monitoring Committee
DNA deoxyribonucleic acid

DSPH (Gilead) Drug Safety and Public Health

ECG electrocardiogram

eCRF electronic case report form
EDC electronic data capture

eg example given ER emergency room

eSAE electronic serious adverse event

ESLD end stage liver disease
ET early termination
EU European Union

EudraCT European Union Drug Regulating Authorities Clinical Trials

FACIT-F Fatigue Index FAS full analysis set

FDA (United States) Food and Drug Administration

FDC fixed-dose combination

FEV1 forced expiratory volume in 1 second

FSH follicle stimulating hormone

g grams

GCP Good Clinical Practice
GGT gamma glutamyl transferase

GI giga

GMR geometric mean ratio

GS-7977 sofosbuvir, formerly PSI-7977

GSI Gilead Sciences, Inc.

GT genotype
h hour
H2 histamine
Hb hemoglobin
HbA1c hemoglobin A1c

HBsAg hepatitis B surface antigen

HBV hepatitis B virus

HCC hepatocellular carcinoma

HCV hepatitis C virus

HDPE high density polyethylene
HIV human immunodeficiency virus

HLGT high-level group term HLT high-level term

HMG-CoA 3-hydroxy-3-methyl-glutaryl coenzyme A

HPF high power field

HRQoL Health Related Quality of Life

IB investigator brochure
ICF informed consent form

ICH International Conference on Harmonization

IEC independent ethics committee

IFN interferon

LH luteinizing hormone

ie in essence

IL28B interleukin-28B gene
IMB intermenstrual bleeding

IMP Investigational Medicinal Product
IND Investigational New Drug (Application)

INR international normalized ratio of prothrombin time

IRB institutional review board

IU International Units
IUD intrauterine device

IUS intrauterine hormone-releasing system

IV intravenous

IWRS interactive web response system

J-GCP Ministerial Ordinance on Good Clinical Practice for Drugs

kg kilogram kPA kilopascal L liter

LAM lactational amenorrhea method

LDL low-density lipoprotein

LDV ledipasvir

LLN lower limit of the normal range LLOQ lower limit of quantification

LLT lower-level term m<sup>2</sup> square meter

MCV mean corpuscular volume or mean cell volume

MELD Model for End Stage Liver Disease

MedDRA Medical Dictionary for Regulatory Activities

mEq milliequivalents mg milligram

MGB minor groove binder MH Mantel-Haenszel

MHLW Ministry of Health, Labour and Welfare

mL milliliter

mm<sup>3</sup> cubic millimeter mmHg millimeters mercury

mmol millimole n number NGM/EE norgestimate/ethinyl estradiol

NS (3/4A/5A/5B) non-structural protein OC hormonal contraceptive **PCR** polymerase chain reaction Peg-IFN pegylated interferon p-glycoprotein P-gp PK

**PMDA** Pharmaceuticals and Medical Devices Agency

pharmacokinetic

**PPIs** proton-pump inhibitors

PR P and R waves (in electrocardiography) PT preferred term or prothrombin time

Q1 quartile 1 Q3 quartile 3 QTc corrected QT

**RAV** resistance-associated variants

**RBC** red blood cell count

**RBV** ribavirin

**RNA** ribonucleic acid

**SADR** serious adverse drug reaction

SAE serious adverse event Scr serum creatinine (mg/dL) SD standard deviation

sec seconds

SF-36 36-Item Short Form Health Survey **SGOT** serum glutamic oxaloacetic transaminase **SGPT** serum glutamic-pyruvic transaminase **SNP** single nucleotide polymorphism

SOC system Organ Class

SOF sofosbuvir, formerly GS-7977 SOP standard operating procedure

STR single tablet regimen

**SUSAR** Suspected Unexpected Serious Adverse Reaction

**SVR** sustained virologic response

SVR12 sustained virologic response 12 weeks after cessation of treatment SVR24 sustained virologic response 24 weeks after cessation of treatment SVR4 sustained virologic response 4 weeks after cessation of treatment

**TEN** toxic epidermal necrolysis

**TIPS** transjugular intrahepatic portosystemic shunt

**TND** target not detected **ULN** upper limit of normal US United States
WBC white blood cell

WPAI Work Productivity and Activity Impairment

VEL velpatasvir

β-hCG β-human chorionic gonadotropin

 $\begin{array}{ll} \mu g & microgram \\ \mu L & microliter \\ \mu mol & micromole \end{array}$ 

# 1. INTRODUCTION

# 1.1. Background

Hepatitis C virus infection is a global health challenge with the estimated number of persons infected ranging from 80 to 150 million worldwide {Gower et al 2014, World Health Organization (WHO) 2016}. Hepatitis C virus has significant genetic (RNA sequence) variability and is classified on this basis into at least 6 genotypes. There is significant geographical variation in the distribution of HCV genotypes. In North America and Europe, genotype 1 HCV infection predominates. In Asia, genotype 1 and 3 HCV infections are the most prevalent. Genotypes 4, 5 and 6 are highly prevalent in Northern Africa, Southern Africa, and Southeast Asia, respectively.

The disease burden of HCV infection is due to progression of chronic liver disease, which can lead to cirrhosis, liver failure, hepatocellular carcinoma (HCC), and death. Globally, 27% of all patients with cirrhosis and 25% of those who develop HCC are attributable to HCV infection {Perz et al 2006}. In addition to having a higher incidence of HCC, patients with chronic HCV infection have a higher incidence and mortality of many types of nonliver cancers including pancreatic, rectal, kidney, non-Hodgkin's lymphoma and lung cancers, compared with the general population {Allison et al 2015}. Curing HCV infection is associated with numerous health benefits including more than 70% reduction in the risk of HCC and a 90% reduction in the risk of liver-related mortality and liver transplantation {Morgan et al 2013, Poynard et al 2002, van der Meer et al 2012, Veldt et al 2007}.

Recently, there has been a transformation in the treatment of HCV infection with the development of direct-acting antivirals (DAAs) targeting viral proteins essential to viral replication. DAA based treatment regimens are generally well tolerated and result in high rates of sustained virologic response at 12 weeks following completion of all treatment (SVR12) across most patient populations {Gilead Sciences Inc 2013, Gilead Sciences Inc 2016a, Gilead Sciences Inc 2016b, Gilead Sciences International Ltd. 2016}. Sofosbuvir (SOF)-based regimens are the most widely prescribed treatments for HCV infection due to the efficacy, tolerability, and simplicity of the dosing regimens. In addition, SOF-based regimens offer the advantages of having relatively few drug-drug interactions, strong concordance between clinical trial and "real world" data, and absence of a requirement for baseline NS5A polymorphism testing {Ioannou et al 2016}. The recent approvals in the US and EU of Epclusa®, a fixed dose combination of SOF and velpatasvir (VEL), are important advancements in HCV drug development as Epclusa® is highly efficacious across all HCV genotypes whereas previously approved regimens were HCV genotype specific {Arias et al 2016, Gilead Sciences Inc 2013, Gilead Sciences Inc 2016a, Gilead Sciences International Ltd 2016, Ioannou et al 2016}

#### 1.1.1. HCV Infection in Japan

With published HCV prevalence estimates from blood-donor and subgroup-based studies on the order of 1-1.9% in Japan {Sievert et al 2011}, it is estimated that there are approximately 1.3-2.4 million people chronically infected with HCV. The highest prevalence rates of HCV

antibodies in first-time blood donor studies have been reported in the 50-59 year (1.8%) and 60-69 year (3.4%) age groups {Tanaka et al 2004}. It is estimated that approximately 15-30% of patients with chronic hepatitis C will go on to develop complications including liver cirrhosis, HCC, and end stage liver disease (ESLD) {Thein et al 2008}. In Japan, HCV genotype 1 and genotype 2 are the predominant genotypes which account for approximately 70% and 30% of chronic infections, respectively {Chung et al 2010}.

# 1.2. Sofosbuvir/Velpatasvir Fixed-Dose Combination

Sofosbuvir (SOF) is a nucleotide analog HCV NS5B polymerase inhibitor. Velpatasvir (VEL) is a pangenotypic HCV NS5A inhibitor.

#### **1.2.1** General Information

Please refer to the Investigator's Brochure (IB) for additional information on SOF/VEL, and the individual components, including:

- InVitro Anti-Hepatitis C Virus Activity
- Nonclinical Pharmacokinetics and In Vitro Metabolism
- Nonclinical Pharmacology and Toxicology
- Clinical Experience

#### 1.3. Information about Ribavirin

Ribavirin (RBV) is a guanosine analogue that inhibits the *in vitro* replication of a wide range of RNA and DNA viruses {MSD K.K. Kudan-kita Chiyoda-ku 2016}. RBV monotherapy has little or no effect on the replication of HCV *in vivo* but can result in normalization of serum ALT activity and improvement in liver histology. RBV is a known teratogen. Furthermore, RBV is known to accumulate intracellularly where it is cleared slowly, and is also excreted in semen. Therefore, extreme care must be taken to avoid pregnancy during RBV therapy and for up to 6 months following completion of treatment. A comprehensive review of RBV is contained in the REBETOL® package insert.

# 1.4. Rationale for This Study

The GS-US-342-4019 study is a Phase 3 multicenter, open-label study evaluating SOF/VEL ± RBV for 12 weeks in subjects with HCV infection and Child-Pugh-Turcotte (CPT) class B or C cirrhosis. Approximately 100 subjects will be enrolled.

SOF/VEL with RBV for 12 weeks is approved in the US and EU (as Epclusa®) for the treatment of HCV infection in patients with decompensated cirrhosis based on the results of the ASTRAL-4 study {Curry et al 2015}. Of the 87 HCV infected subjects treated with SOF/VEL and RBV for 12 weeks in the ASTRAL-4 study, 82 (94%) achieved SVR12 (ranging from

85% in GT3 to 100% in GT2 and GT4). In GT1, the SVR12 rates were 94% and 100% in GT1a and GT1b, respectively.

Of the 90 subjects treated with SOF/VEL for 12 weeks, 75 (83%) achieved SVR12 (ranging from 50% in GT3 to 100% in GT2 and GT4 subjects). The majority of subjects were GT1 with SVR rates of 88% in GT1a and 89% in GT1b. The majority of Japanese patients with chronic HCV are elderly (average age  $\sim$  70 years), are more likely to be treatment-experienced, and have progressive liver disease. Comorbid conditions (e.g., diabetes and cardiovascular disease) are common in this population and pose challenges to the use of RBV therapy. Therefore, SOF/VEL will be evaluated both with and without RBV.

# 1.5. Rationale for Dose Selection of SOF/VEL

Subjects in this study will be administered SOF/VEL, a co-formulation of SOF 400 mg and VEL 100 mg that is approved in the US, EU, and other regions as Epclusa<sup>®</sup> for the treatment of HCV infection in adults.

In the Phase 3 ASTRAL 1-3 studies, treatment of HCV infected subjects infected without cirrhosis or with compensated cirrhosis for 12 weeks with SOF/VEL was well tolerated and resulted in high SVR12 rates. In the ASTRAL-4 study, treatment of HCV-infected subjects with decompensated Child Pugh Turcotte class B cirrhosis with SOF/VEL and ribavirin for 12 weeks was well tolerated and resulted in high SVR12 rates across all HCV genotypes evaluated.

Based on these data, the results of Phase 1 studies in subjects with hepatic impairment and population PK analyses from studies of HCV-infected subjects, no dose adjustment of SOF/VEL is recommended in patients with CPT C cirrhosis. Refer to the SOF/VEL Investigator's Brochure for additional information.

#### 1.6. Rationale for Dose Selection of Ribavirin

Data from the ASTRAL-4 and SOLAR studies support the use of different starting doses of RBV based on subject's CPT class at Screening so that subjects with CPT B cirrhosis will start at 600-1000 mg daily based on weight, whereas subjects with CPT C cirrhosis will start at 600 mg daily.

The SOLAR-1 and SOLAR -2 studies evaluated ledipasvir (LDV)/SOF and RBV 600mg for 12 or 24 weeks in pre and posttransplant subjects with advanced liver disease including subjects with decompensated cirrhosis {Charlton et al 2015, Manns et al 2016}. In these studies, treatment of subjects with CPT C cirrhosis with LDV/SOF and RBV 600mg for 12 or 24 weeks was well tolerated and resulted in high SVR12 rates. Based on the SOLAR-1 and SOLAR-2 data, the US PI and EU SmPC for Harvoni recommended a 600 mg starting dose of RBV in HCV infected patients with decompensated cirrhosis {Gilead Sciences Inc 2016b, Gilead Sciences International Ltd. 2016}.

The ASTRAL-4 study evaluated the safety and efficacy of SOF/VEL with and without RBV (1000-1200 mg daily weight-based, per the RBV US PI and SmPC) per the RBV US PI and

SmPC for 12 weeks and SOF/VEL for 24 weeks in patients with decompensated cirrhosis. Of 87 subjects treated with SOF/VEL and RBV for 12 weeks, 77 (89%) had CPT B cirrhosis and 4 (5%) had CPT C cirrhosis at baseline. RBV dose reduction was required by approximately one third of subjects with CPT B cirrhosis compared with 3 of 4 subjects with CPT C cirrhosis suggesting that weight based (1000-1200 mg) RBV dosing was less tolerated in patients with CPT C cirrhosis compared with patients with CPT B cirrhosis.

# 1.7. Risk/Benefit Assessment for the Study

This study will provide information of the safety and efficacy of the combination of SOF/VEL with or without RBV for 12 weeks in Japanese patients with decompensated cirrhosis.

The safety profile of SOF/VEL has been established in 3126 subjects, including 1558 subjects in the Phase 3 studies, 802 in the Phase 2 studies, 499 in the Phase 1 studies, and 267 subjects with decompensated cirrhosis in the Phase 3 Study GS-US-342-1137 (ASTRAL-4). No clinical safety issues specifically related to the combination of SOF/VEL have been identified to date. Overall, SOF/VEL plus RBV for 12 weeks was safe and well tolerated in patients with CPT B cirrhosis.

During the conduct of the study, the sponsor will perform ongoing safety review and a Data Monitoring Committee (DMC) will meet to review safety data.

In summary, safety and efficacy of SOF/VEL with and without RBV for 12 weeks has been evaluated in subjects with CPT B cirrhosis in overseas studies. This study will be the first to evaluate SOF/VEL with and without RBV in Japanese patients with decompensated cirrhosis.

# 1.8. Compliance

This study will be conducted in accordance with ICH Good Clinical Practice (GCP), and J-GCP (Ministerial Ordinance on Good Clinical Practice for Drugs), and all applicable regulatory requirements, including archiving of essential documents.

# 2. OBJECTIVES

The primary objectives of this study are:

- To evaluate the antiviral efficacy of therapy with sofosbuvir/velpatasvir (SOF/VEL)
  fixed-dose combination (FDC) with or without ribavirin for 12 weeks as measured by the
  proportion of subjects with sustained virologic response 12 weeks after cessation of treatment
  (SVR12)
- To evaluate the safety and tolerability of each treatment regimen

The secondary objectives of this study are:

- To determine the proportion of subjects who attain SVR at 4 and 24 weeks after cessation of treatment (SVR4 and SVR24)
- To evaluate the proportion of subjects with virologic failure
- To evaluate therapeutic efficacy as measured by the change of CPT score and MELD score
- To evaluate the kinetics of circulating HCV RNA during treatment and after cessation of treatment
- To evaluate the emergence of viral resistance to SOF and VEL during treatment and after cessation of treatment

The exploratory objectives of this study are:



# 3. STUDY DESIGN

# 3.1. Study Design

This is a multicenter, randomized, open-label study evaluating the efficacy and safety of  $SOF/VEL \pm RBV$  for 12 weeks in subjects with chronic HCV infection with decompensated cirrhosis.

Initially only subjects with CPT B cirrhosis at Screening (score 7-9) will be enrolled. Enrollment of subjects with CPT C cirrhosis at Screening (score 10-12) will begin after the DMC has reviewed accumulated safety data from the first 20 subjects through 4 weeks of treatment (or early treatment discontinuation) and concluded that these data support enrollment of subjects with CPT C cirrhosis.

# 3.2. Study Treatments

Approximately 100 subjects will be randomized (1:1) to one of the following two treatment groups:

- SOF/VEL (400/100 mg) for 12 weeks (n=50)
- SOF/VEL (400/100 mg) with RBV for 12 weeks (n=50)

Randomization will be stratified by Child-Pugh-Turcotte (CPT) class at Screening (CPT B/ CPT C) and HCV genotype (genotype 1/ non-genotype 1). For the purposes of randomization, a subject with non-definitive or mixed HCV genotype results by central laboratory analysis will be considered non-genotype 1. At least 15 subjects will have non-genotype 1 HCV infection. Approximately 10% of subjects will have CPT C (score 10-12) decompensated cirrhosis.

#### 3.3. Duration of Treatment

Subjects will be treated for 12 weeks.

The total time to complete all study visits is approximately 40 weeks (42 weeks for those requiring an extension of the Screening period):

- 28 days (4 weeks) screening period
- 12 weeks study treatment period
- 24 weeks posttreatment period

# 3.4. Stopping Rules and Discontinuation Criteria

If a subject discontinues study dosing (for example, as a result of an adverse event [AE]), every attempt should be made to keep the subject in the study and continue to perform the required

study-related follow-up procedures (see Section 6.5). If this is not possible or acceptable to the subject or investigator, the subject may be withdrawn from the study.

There is no option for SOF/VEL dose reduction. If SOF/VEL is withheld due to toxicity, the subject must also discontinue RBV treatment (if applicable). Subjects that require discontinuation of only RBV for RBV-related events should continue with SOF/VEL for the remainder of the treatment period and complete all scheduled study visits.

Subjects who permanently discontinue SOF/VEL should complete an Early Termination (ET) visit. For subjects who have completed an ET visit, the posttreatment Week 4, 12, and 24 visits will be completed after the last dose of any of the study drugs. When medically feasible, the medical monitor must be consulted prior to subject discontinuation.

Study drug must be discontinued in the following instances:

- Unacceptable toxicity, as defined in Section 3.4.1, or toxicity that, in the judgment of the investigator, compromises the ability to continue study-specific procedures or is considered to not be in the subject's best interest
- It is expected that some subjects will have progression of their liver disease during the study. The decision to continue such subjects on treatment will be made by the investigator based on assessment of the risk/benefit for the individual patient
- Virologic failure (as defined in Section 3.4.2)
- Pregnancy of female subject (refer to Appendix 4)
  - In the event that the female partner of a male subject receiving SOF/VEL+RBV becomes pregnant, the subject must discontinue RBV but may continue treatment with SOF/VEL (refer to Section 7.5.1)
- Significant protocol violation including non-compliance with study assessments
- Subject request to discontinue for any reason; it is important to determine whether the withdrawal of consent is primarily due to an AE, lack of efficacy, or other reason
- Discontinuation of the study at the request of Gilead, regulatory agency or an Institutional Review Board (IRB)/Independent Ethics Committee (IEC)

#### 3.4.1. Toxicity-Based Stopping Criteria

Subjects who meet any of the following laboratory or adverse event criteria must stop treatment with SOF/VEL:

- Confirmed total bilirubin > 3x Day 1 or nadir and ALT and/or AST > 3x Day 1 or nadir
- Elevation of alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) > 10x Day 1 or nadir, confirmed by immediate repeat testing

- Any Grade 3 or greater rash associated with constitutional symptoms
- Any Grade 4 adverse event assessed as related to administration of SOF/VEL

# 3.4.2. Virologic Response-Based Treatment Stopping Criteria

The following on-treatment Virologic Response-based Treatment Stopping Criteria will be utilized:

- Confirmed HCV RNA ≥ LLOQ after 2 consecutive HCV RNA < LLOQ</li>
- Confirmed > 1 log<sub>10</sub> increase in HCV RNA from nadir
- HCV RNA ≥ LLOQ through 8 weeks of treatment

Confirmation should be performed as soon as possible and must occur no later than 2 weeks after an initial observation indicating virologic failure during the on-treatment phase.





PPD

# 4. SUBJECT POPULATION

# 4.1. Number of Subjects and Subject Selection

Approximately 100 chronic HCV infected, male and non-pregnant female subjects, ages 20 years or older with CPT class B or C cirrhosis at Screening will be enrolled in this study.

In order to manage the total study enrollment, Gilead Sciences, Inc., at its sole discretion, may suspend screening and/or enrollment at any site or study-wide at any time.

#### 4.2. Inclusion Criteria

Subjects must meet *all* of the following inclusion criteria to be eligible for participation in this study.

- 1) Willing and able to provide written informed consent
- 2) Male or female, age  $\geq$  20 years at Screening
- 3) Body weight  $\geq$  40 kg at Screening
- 4) Quantifiable HCV RNA at Screening
- 5) Chronic HCV infection (≥ 6 months prior to Screening) documented by prior medical history or liver biopsy
- 6) Confirmation of cirrhosis by any one of the following methods:
  - a) Liver biopsy showing cirrhosis (eg. Metavir score = 4 or Ishak score  $\geq 5$ )
  - b) Fibroscan showing cirrhosis or results > 12.5 kPa
  - c) FibroTest® score of > 0.75 (only in the absence of liver biopsy or availability of Fibroscan)
- 7) CPT score 7 to 12, inclusive, at Screening as determined using laboratory values from the central laboratory, and at Day 1 (before dosing) using laboratory values from the local laboratory
- 8) Liver imaging (eg, ultrasound or CT scan, at the discretion of the investigator) performed within 4 months of Day 1 to exclude hepatocellular carcinoma (HCC)
- 9) If treatment-experienced, the most recent HCV treatment must have been completed at least 8 weeks prior to Screening
- 10) If listed for liver transplant, Day 1 is expected to be at least 12 weeks prior to transplant.

- 11) Females of childbearing potential (as defined in Appendix 4) must have a negative serum pregnancy test at Screening and a negative urine pregnancy test on Day 1 prior to randomization.
- 12) Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception as described in Appendix 4.
- 13) Female subjects must agree to refrain from egg donation and in vitro fertilization during treatment until at least 6 months after the last dose of RBV or 30 days after the last dose SOF/VEL, whichever occurs last.
- 14) Male subjects must agree to refrain from sperm donation from the date of screening until at least 6 months after the last dose of RBV or 30 days after the last dose SOF/VEL, whichever occurs last
- 15) Lactating females must agree to discontinue nursing before the study drugs are administered and through at least 12 weeks after the last dose of any study drug.
- 16) Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments, including all required posttreatment visits.

#### 4.3. Exclusion Criteria

Subjects who meet any of the following exclusion criteria are not to be enrolled in this study.

- 1) Current or prior history of any of the following:
  - a) Clinically significant illness or currently under evaluation for a potentially clinically significant illness (other than HCV or co-morbidities associated with advanced liver disease except as noted below) or any other major medical disorder that may interfere with subject treatment, assessment or compliance with the protocol.
  - b) Gastrointestinal disorder or postoperative condition that could interfere with the absorption of the study drugs
  - c) Difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
  - d) Solid organ transplantation
  - e) Significant pulmonary disease
  - f) Unstable cardiac disease or significant cardiac event within one year prior to Screening
  - g) Porphyria

- h) Clinically significant hemoglobinopathy (e.g., thalassemia, sickle cell anemia)
- i) Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 2 years prior to Screening
- j) Malignancy, other than hepatocellular carcinoma, within the 5 years prior to screening with the exception of specific cancers that have been cured by surgical resection (basal cell skin cancer, etc.). Subjects under evaluation for possible malignancy are not eligible.
- k) Hepatocellular carcinoma within 2 years prior to Screening. Subjects with a history of HCC that was curatively treated with either surgical resection or radiofrequency ablation (RFA), with the end of treatment occurring at least 2 years prior to Screening, are eligible for enrollment.
- 1) Recurrence of hepatocellular carcinoma after curative treatment
- m) Significant drug allergy (such as anaphylaxis or hepatotoxicity)
- n) Hepatopulmonary syndrome
- o) Hepatorenal syndrome
- 2) Infection with human immunodeficiency virus (HIV) at Screening
- 3) Hepatitis B virus (HBV) surface antigen positive at Screening
- 4) Screening ECG with clinically significant abnormalities
- 5) Prior exposure to any HCV NS5A inhibitor
- 6) Use of GM-CSF, epoetin alfa or other hematopoietic stimulating agents within 2 weeks of Screening
- 7) Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, autoimmune hepatitis, Wilson's disease, α-1-antitrypsin deficiency, alcoholic liver disease, non-alcoholic steatohepatitis, or toxin exposures)
- 8) Pregnant or nursing female or male with pregnant female partner
- 9) Women who wish to become pregnant or males with female partners who wish to become pregnant during study treatment and through 6 months after the last dose of RBV or 30 days after the last dose SOF/VEL whichever comes last
- 10) Chronic use of systemically administered immunosuppressive agents (eg, prednisone equivalent > 10 mg/day)
- 11) Active spontaneous bacterial peritonitis at Screening


- 12) Infection requiring systemic antibiotics at the time of Screening
- 13) Evidence of fibrosing cholestatic hepatitis
- 14) Life threatening SAE during Screening
- 15) Active variceal bleeding within 6 months of Screening
- 16) Prior placement of a portosystemic shunt (such as TIPS)
- 17) Subjects with any of the following laboratory parameters at Screening:
  - a) Hemoglobin (Hb) < 11 g/dL for female subjects; Hb < 12 g/dL for male subjects
  - b) Platelets  $< 50,000/\text{mm}^3$
  - c) Neutrophils <1000/mm<sup>3</sup>
  - d) ALT, AST, or alkaline phosphatase  $\geq 10 \text{ x ULN}$
  - e) Sodium <125 mEq/L
  - f) Total bilirubin > 10 mg/dL
  - g) Creatinine clearance ( $CL_{cr}$ ) < 50 mL/min as calculated by the Cockcroft-Gault equation using actual body weight {Cockcroft et al 1976}; ideal body weight may be used on a case-by-case basis when approved by the Medical Monitor.
- 18) Donation or loss of more than 400 mL of blood within 2 months prior to Day 1
- 19) Participation in a clinical study with an investigational drug or biologic within 1 month prior to Screening
- 20) Any contraindication to RBV therapy, per the approved package insert, with the exception of serious hepatic dysfunction
- 21) Any prohibited medications as described in Section 5.6
- 22) Known hypersensitivity to ribavirin, velpatasvir, sofosbuvir, or the metabolites or formulation excipients
- 23) Known contraindication to sofosbuvir per the approved package insert


#### 5. INVESTIGATIONAL MEDICINAL PRODUCTS

# 5.1. Randomization, Blinding and Treatment Codes

This is a multicenter, randomized, open-label study in subjects with chronic HCV infection with decompensated cirrhosis. No blinding is required.

Approximately 100 subjects will be randomized (1:1) to one of the following two groups:

- SOF/VEL (400/100 mg) for 12 weeks (n=50)
- SOF/VEL (400/100 mg) with RBV for 12 weeks (n=50)

Randomization will be stratified by Child-Pugh-Turcotte (CPT) class (CPT B/ CPT C) at Screening and HCV genotype (genotype 1/ non-genotype 1). Any non-definitive or mixed HCV genotype results will be considered non-genotype 1 for randomization purposes. At least 15 subjects will have non-genotype 1 HCV infection. Approximately 10% of subjects will have CPT C (score 10-12) decompensated cirrhosis.

Initially only subjects with CPT B cirrhosis at Screening (score 7-9) will be enrolled. Enrollment of subjects with CPT C cirrhosis at Screening (score 10-12) will begin after the DMC has reviewed accumulated safety data from the first 20 subjects through 4 weeks of treatment (or early treatment discontinuation) and concluded that these data support enrollment of subjects with CPT C cirrhosis.

# 5.2. Description and Handling of SOF/VEL FDC

#### **5.2.1.** Formulation

The SOF/VEL (400/100 mg) tablets are pink, diamond-shaped, film-coated tablets, debossed with "GSI" on one side and "7916" on the other side. In addition to the active ingredients, the SOF/VEL tablets contain copovidone, microcrystalline cellulose, croscarmellose sodium, magnesium stearate, polyvinyl alcohol, titanium dioxide, polyethylene glycol, talc, and iron oxide red.

# 5.2.2. SOF/VEL FDC Packaging and Labeling

SOF/VEL (400/100 mg) tablets are packaged in white, high density polyethylene (HDPE) bottles. Each bottle contains 28 tablets and polyester packing material. Each bottle is enclosed with a white, continuous thread, child-resistant screw cap with an induction-sealed, aluminum-faced liner.

SOF/VEL bottles to be distributed to centers in Japan shall be labeled for clinical use to meet applicable requirements of the J-GCP (Ministerial Ordinance on Good Clinical Practice for Drugs).

# **5.2.3. SOF/VEL FDC Storage and Handling**

SOF/VEL FDC tablets should be stored at controlled room temperature until required for administration. Controlled room temperature is defined as 25°C (77 °F); excursions are permitted between 15°C and 30°C (59°F to 86°F).

All drug products should be stored in a securely locked area, accessible only to authorized site personnel. To ensure the stability of the study drugs and to ensure proper product identification, the drug product should not be stored in a container other than the container in which they are supplied. Consideration should be given to handling, preparation, and disposal through measures that minimize drug contact with the body. Appropriate precautions should be followed to avoid direct eye contact or exposure through inhalation when handling SOF/VEL tablets.

Sufficient quantities of SOF/VEL FDC tablets to complete the entire study will be shipped to the investigator or qualified designee from the Gilead Clinical Supply Management Team (or its designee).

# **5.2.4.** Dosage and Administration of SOF/VEL FDC

SOF/VEL tablet is to be administered once daily with or without food. Each subject must be given instructions to maintain approximately the same daily dosing interval between study drugs doses.

If a subject does not take the SOF/VEL FDC dose at the usual time, it may be taken up to 18 hours later; however, no more than one tablet should be taken on any calendar day. The subject should resume the standing dosing schedule on the next day.

Study drugs should not be cut or split. SOF/VEL FDC tablets will be provided by Gilead Sciences for all subjects.

# 5.3. Description and Handling of Ribavirin (RBV)

#### **5.3.1.** Formulation

RBV will be provided in the course of this study as REBETOL® capsules (MSD K.K.). REBETOL® capsules are white opaque hard capsules. Each capsule contains 200 mg of ribavirin. Information regarding commercially available REBETOL® capsules can be found in the current prescribing information {MSD K.K. Kudan-kita Chiyoda-ku 2016}.

#### 5.3.2. RBV Packaging and Labeling

REBETOL<sup>®</sup> capsules are packaged in blister packaging of 140 capsules. The RBV package shall be labeled for clinical use to meet all applicable requirements of the J-GCP (Ministerial Ordinance on Good Clinical Practice for Drugs).

# 5.3.3. RBV Storage and Handling

Information regarding commercially available REBETOL® capsules can be found in the current prescribing information.

All drug products should be stored in a securely locked area, accessible only to authorized site personnel. To ensure the stability of the study drug and to ensure proper product identification, the drug product should not be stored in a container other than the container in which they are supplied. Consideration should be given to handling, preparation, and disposal through measures that minimize drug contact with the body. Appropriate precautions should be followed to avoid direct eye contact or exposure through inhalation when handling RBV.

# **5.3.4.** Dosage and Administration of RBV

For subjects with CPT B cirrhosis at Screening, RBV dosage will be based on weight. Subjects with CPT C cirrhosis at Screening will be administered 600 mg in a divided daily dose. See Table 5-1 below.

| Table 5-1. | Dosing and Administration of RBV |
|------------|----------------------------------|
|------------|----------------------------------|

| | | Ribavirin dosage | | |
|---|---|---|---|---|
| CPT Class | Body Weight at<br>Day 1 | Daily dosage | After morning meal | After evening meal |
| СРТ В | ≤ 60 kg | 600 mg | 200 mg | 400 mg |
| | > 60 kg to ≤ 80 kg | 800 mg | 400 mg | 400 mg |
| | > 80 kg | 1,000 mg | 400 mg | 600 mg |
| CPT C | - | 600 mg | 200 mg | 400 mg |

Recommendations for RBV dose modification or discontinuation are in Section 7.5.1.

RBV should be dosed with food and SOF/VEL when appropriate.

RBV capsule (200 mg) will be supplied by Gilead Sciences for all applicable subjects.

#### 5.4. Co-administration of SOF/VEL and RBV

For <u>morning doses</u>, subjects will be instructed to take study drugs <u>with food</u> as follows:

- One SOF/VEL FDC Tablet: contains 400 mg of SOF and 100 mg of VEL
- RBV as per Table 5-1

For <u>evening doses</u>, subjects will be instructed to take study drug <u>with food</u> as follows:

• RBV as per Table 5-1

If a subject does not take the SOF/VEL dose at the usual time, it may be taken up to 18 hours later; however, no more than one tablet should be taken on any calendar day. The subject should resume the standing dosing schedule on the next day.

RBV should be administered as a divided daily dose (i.e., morning and evening) per Table 5-1. If the subject misses a dose of RBV and remembers the same day, the missed dose should be taken as soon as possible. However, if the subject missed taking the morning dose with lunch or if more than 6 hours have passed since the usual morning dose time, the subject should only take the prescribed evening dose of RBV. Subjects should be instructed <u>not</u> to take his/her morning and evening doses of RBV at the same time.

Study drugs should not be cut or split. No food restrictions apply to SOF/VEL; however, SOF/VEL should be taken with the morning dose of RBV which is taken with food.

# 5.5. Study Drug Adherence and Drug Accountability

Subjects must be instructed to bring back all study drug(s) in the original container at every study visit after Day 1 through the end of treatment.

Study drug(s) will be reconciled using medication pill count at every post-Day 1 visit by the investigator or designee (ie, pharmacist) in order to monitor the subject's adherence with the study drug(s).

#### 5.6. Prior and Concomitant Medications

All concomitant medications taken within 30 days prior to Screening, up to and including 30 days after the last dose of study drug, need to be recorded in the source documents and eCRF (including all blood products). In addition, records of concomitant medications for ascites and hepatic encephalopathy taken through posttreatment Week 24 will be collected in the eCRF.

Investigational agents or devices for any indication are prohibited from 28 days prior to the Day 1 visit through the end of study drug dosing.

Concomitant use of certain medications or herbal/natural supplements (such as moderate to potent inducers of drug transporters or metabolizing enzymes, eg, P-gp, CYP2B6, CYP2C8, or CYP3A) with the study drug may result in pharmacokinetic interactions resulting in increases or decreases in exposure of the study drug or these medications.

Table 5-2 below contains examples of medications that are prohibited from 21 days prior to Day 1 through the end of treatment and those medications which may be used with caution. The use of amiodarone is prohibited from 60 days prior to Day 1 through the end of treatment.

Additionally, investigators should refer to the product/package inserts of other medications for age-related recommendations or contraindications related to their use.

Table 5-2. Disallowed and Concomitant Medications to be Used with Caution

| Drug Class | Agents Disallowed | <b>Use with Caution</b> |
|---|---|---|
| Acid Reducing Agents <sup>a</sup> | | Proton- Pump Inhibitors, H2-Receptor<br>Antagonists, Antacids |
| Anticonvulsants <sup>b</sup> | Phenytoin, Carbamazepine, Phenobarbital,<br>Oxcarbazepine | |
| Antimycobacterials <sup>b</sup> | Rifampicin, Rifabutin, Rifapentine <sup>g</sup> | |
| Cardiac Medications <sup>c</sup> | Amiodarone <sup>d</sup> | Digoxin <sup>e</sup> |
| Herbal/Natural<br>Supplements <sup>b</sup> | St. John's Wort, Echinacea, Milk thistle (i.e., silymarin), Chinese herb sho-saiko-to (or Xiao-Shai-Hu-Tang) | |
| HMG-CoA Reductase<br>Inhibitors <sup>f</sup> | | Rosuvastatin (≤10 mg/day) <sup>f</sup> , Atorvastatin |
| Other | Bosentan <sup>b</sup> , Modafinil <sup>b</sup> , Sulfasalazine <sup>c</sup> , , Methotrexate <sup>c</sup> | |

a Proton pump inhibitor (PPI) doses comparable with omeprazole 20mg can be administered with SOF/VEL when SOF/VEL is administered with food. H2-receptor antagonists must not exceed a dose of 40 mg famotidine or equivalent and can be taken simultaneously with SOF/VEL and/or staggered by 12 hours. Antacids that directly neutralize stomach acid may not be taken within 4 hours (before or after) of SOF/VEL administration.

- b May result in a decrease in the concentration of study drugs.
- c May result in an increase in the concentration of study drugs and/or concomitant medications
- d May result in symptomatic bradycardia. Mechanism is not currently known. The use of amiodarone is prohibited from 60 days prior to Day 1 through the end of treatment
- e Monitor for signs and symptoms of digoxin toxicity.
- f Use with SOF/VEL may result in an increase in the concentration of HMG-CoA Reductase Inhibitor, rosuvastatin. Monitor for signs and symptoms of muscle weakness or myopathy, including rhabdomyolysis.
- g Unapproved in Japan

Medications for disease conditions **excluded** from the protocol (eg, HIV infection) are not listed under this Concomitant Medication section and are disallowed in the study.

Should subjects have a need to initiate treatment with any excluded concomitant medication, the Medical Monitor must be consulted prior to initiation of the new medication. In instances where an excluded medication is initiated prior to discussion with the Sponsor, the Investigator must notify Gilead as soon as he/she is aware of the use of the excluded medication.

# **Colony Stimulating Agents**

Potential subjects may not be treated with colony stimulating agents (CSA) within **2 weeks prior to Screening and through Day 1** to elevate hematology laboratory parameters to facilitate entry into the study. Use during the study is allowed as clinically indicated.

# 5.7. Accountability for Study Drug

The investigator or designee (ie, pharmacist) is responsible for ensuring adequate accountability of all used and unused study drugs. This includes acknowledgement of receipt of each shipment of study drugs (quantity and condition). All used and unused study drugs dispensed to subjects must be returned to the site

SOF/VEL and RBV accountability records will be provided to each study site to:

- Record the lot number, expiration date (if necessary)
- Record the date received and quantity of study drugs kits
- Record the date, subject number, the study drugs kit number dispensed
- Record the date, quantity of used and unused study drugs returned, along with the initials of the person recording the information.

# 5.7.1. Study Drug Return or Disposal

Refer to Section 9.1.7 for information on return and disposal of study drugs.

#### 6. STUDY PROCEDURES

The study procedures to be conducted for each subject enrolled in the study are presented in tabular form in Appendix 2 and described in the text that follows

The investigator must document any deviation from protocol procedures and notify the sponsor or contract research organization (CRO).

# 6.1. Screening Visit

Screening assessments will be completed within 28 days of the Day 1 visit. The screening window can be extended up to 42 days for subjects for extenuating circumstances with sponsor approval. A single retest of screening labs is permitted only if there is reason to believe the retest value will be within accepted parameters if the initial value was either due to a sample processing error or due to an extenuating circumstance such as intercurrent infection.

The following procedures will be performed and documented:

Obtain written informed consent



- Determine inclusion and exclusion eligibility
- Obtain medical history (refer to Section 6.8.2), including:
  - Hepatitis C treatment history, if applicable
    - Regimen(s)
    - Dates of previous treatment(s)
    - Response to previous treatment (ie, nonresponder, relapse, discontinuation including reason)
- Perform complete physical examination (refer to Section 6.8.3)
- Obtain height and weight
- Obtain vital signs (refer to Section 6.8.4)
- Perform 12-Lead ECG (refer to Section 6.8.5)
- Record any serious adverse events and all adverse events related to protocol mandated procedures occurring after signing of the consent form
- Obtain details of concomitant medications
- Liver Disease Assessment
  - Liver biopsy and/or Fibroscan results (if available)
  - Assess presence and severity of ascites and hepatic encephalopathy for CPT score (refer to Section 6.8.7)
  - Diagnostic imaging (eg, ultrasound or CT scan, at the discretion of the investigator) should be performed to exclude the presence of hepatocellular carcinoma (HCC). Imaging must have been performed within 4 months of Day 1.
- Obtain blood samples for tests (approximately 30 mL of blood will be drawn):
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Serum β-hCG pregnancy test for females of childbearing potential only
  - HCV Genotype
  - HCV antibody, HIV antibody, HBV surface antigen (HBsAg), HBV surface antibody (HBsAb), HBV core antibody (HBcAb)
  - Fibrotest<sup>®</sup>
- Obtain urine sample for:
  - Urinalysis

A CPT Score Confirmation Form will be required to be submitted and reviewed by the Medical Monitor prior to randomization on Day 1. Subjects meeting all of the inclusion criteria and none of the exclusion criteria will return to the clinic for randomization into the study, upon confirmation of CPT score.

From the time of obtaining informed consent through the first administration of study drugs, record all serious adverse events (SAEs), as well as any adverse events related to protocol-mandated procedures on the adverse events case report form (eCRF). All other untoward medical occurrences observed during the screening period, including exacerbation or changes in medical history are to be captured on the medical history eCRF. See Section 7 Adverse Events and Toxicity Management for additional details.

## 6.1.1. Day 1 Assessments

The following Day 1 tests and procedures must be performed prior to enrollment and dosing/dispensation of study drugs:

- Determine inclusion and exclusion eligibility (refer to Sections 4.1 and 4.2)
  - Confirm CPT score is 7-12 using laboratory data from the local laboratory (refer to Section 6.8.7)
- Subject completes Health Related Quality of Life (HRQoL) surveys (refer to Section 6.8.6)
- Perform complete physical examination (refer to Section 6.8.3)
- Obtain weight
- Obtain vital signs (refer to Section 6.8.4)
- Assessment of AEs and concomitant medications
- Conduct pregnancy prevention counseling
- Perform 12-Lead ECG (refer to Section 6.8.5)
- Obtain blood samples for tests (approximately 30 mL of blood will be drawn for required tests):
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral RNA Sequencing / Phenotyping Sample
  - IL28B Genotype
  - Archive plasma sample (for subjects who have consented) (an additional 12 mL of blood will be drawn)
  - Single genomic sample (for subjects who have consented) (an additional 6 mL of blood will be drawn)
- Obtain urine sample for:
  - Pregnancy test for females of childbearing potential only

## 6.2. Study Drug Administration

An Interactive Web Response System (IWRS) will be employed to manage subject enrollment, randomization, and treatment assignment. Randomization stratification factors are described in Section 5.1.

When ready to administer study drugs to the subject:

- Dispense study drugs as directed by the IWRS
- Instruct the subject on the packaging, storage, and administration of study drugs
- Instruct the subject on how to complete the subject diary
- Observe the subject taking the first dose of study drugs. The subject should take the study drugs with food.

# 6.3. Close Monitoring During Early Phase of Treatment for Subjects with CPT C Cirrhosis

Subjects with CPT C cirrhosis at Screening should be monitored closely during treatment with SOF/VEL ± RBV. The extent and duration of monitoring is at the discretion of the Investigator, based on assessment of each individual subject, but may include daily contact with subject (or subject's family) or in-patient hospitalization. Proximity of subject's residence to the investigator's institution should be taken into consideration. The objective of this close monitoring is to facilitate prompt communication and response to adverse events that may occur.

## 6.4. Treatment Assessments (± 3 days)

On-treatment visits will be performed at the end of Weeks 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, and 12 for all subjects.

Study drugs will be reconciled at every post-Day 1 visit by the investigator or designee (ie pharmacist) in order to monitor the subject's adherence with the study drugs.

## 6.4.1. Weeks 1, 3, 5, 6, 7, 9, 10, and 11 ( $\pm$ 3 days)

The following procedures/assessments are to be completed at the end of Weeks 1, 3, 5, 6, 7, 9, 10, and 11:

- Perform complete physical examination (refer to Section 6.8.3)
- Obtain weight
- Obtain vital signs (refer to Section 6.8.4)
- Assessment of AEs and concomitant medications
- Assess adherence with study drug dosing regimen including pill count

## 6.4.2. Week 2 ( $\pm$ 3 days)

The following procedures/assessments are to be completed at the end of Week 2:

- Perform complete physical examination (refer to Section 6.8.3)
- Obtain weight
- Obtain vital signs (refer to Section 6.8.4)
- Assessment of AEs and concomitant medications
- Assess adherence with study drug dosing regimen including pill count
- Obtain blood samples for tests (approximately 40 mL of blood will be drawn total):
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral RNA Sequencing / Phenotyping Sample
  - HBV DNA Sample
  - Single PK sample

#### 6.4.3. Weeks 4 and 8 ( $\pm$ 3 days)

The following procedures/assessments are to be completed at the end of Weeks 4 and 8:

- Perform complete physical examination (refer to Section 6.8.3)
- Obtain weight
- Obtain vital signs (refer to Section 6.8.4)
- Assessment of AEs and concomitant medications
- Assess presence and severity of ascites and hepatic encephalopathy for CPT score (refer to Section 6.8.7)
- Pregnancy prevention counseling

- Assess adherence with study drug dosing regimen including pill count
- Dispense study drugs as directed by the IWRS
- Obtain blood samples for tests (approximately 40 mL of blood will be drawn for required tests):
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral RNA Sequencing / Phenotyping Sample
  - HBV DNA Sample
  - Single PK sample
- Obtain urine sample for:
  - Pregnancy test for females of childbearing potential only

## 6.4.4. Week 12 ( $\pm$ 3 days)

The following procedures/assessments are to be completed at the end of Week 12:

- Subject completes Health Related Quality of Life (HRQoL) surveys (refer to Section 6.8.6)
- Perform complete physical examination (refer to Section 6.8.3)
- Obtain weight
- Obtain vital signs (refer to Section 6.8.4)
- Assessment of AEs and concomitant medications
- Assess presence and severity of ascites and hepatic encephalopathy for CPT score (refer to Section 6.8.7)
- Conduct pregnancy prevention counseling
- Assess adherence with study drug dosing regimen including pill count
- Collect any remaining study drug from the subject

- Obtain blood samples for tests (approximately 40 mL of blood will be drawn for all required tests):
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral RNA Sequencing / Phenotyping Sample
  - HBV DNA Sample
  - Single PK sample
  - Archive plasma sample (for subjects who have consented) (an additional 12 mL of blood will be drawn)
- Obtain urine sample for:
  - Pregnancy test for females of childbearing potential only

#### 6.5. Posttreatment Assessments ( $\pm$ 5 days)

The posttreatment Week 4, 12, and 24 visits should be timed from the date of last administration of any study drugs for all subjects, regardless of whether they are a virologic failure or discontinued study drugs early.

## 6.5.1. Posttreatment Week 4 ( $\pm$ 5 days)

The following procedures/assessments are to be completed for all subjects, 4 weeks after taking the last dose of study drug:

- Perform complete physical examination (refer to Section 6.8.3)
- Obtain weight
- Obtain vital signs (refer to Section 6.8.4)
- Assessment of AEs and concomitant medications
- Assess presence and severity of ascites and hepatic encephalopathy for CPT score (refer to Section 6.8.7)
- Conduct pregnancy prevention counseling

- Obtain blood samples for tests (approximately 35 mL of blood will be drawn total):
  - Hematology
  - Chemistry
  - Coagulation Tests
  - HCV RNA
  - Viral RNA Sequencing / Phenotyping Sample
  - HBV DNA Sample
- Obtain urine sample for:
  - Pregnancy test for females of childbearing potential only (refer to Section 6.8.12)

## 6.5.2. Posttreatment Week 12 ( $\pm$ 5 days)

The following procedures/assessments are to be completed for all subjects, 12 weeks after taking the last dose of study drug:

- Subject completes Health Related Quality of Life (HRQoL) surveys (refer to Section 6.8.6)
- Perform complete physical examination (refer to Section 6.8.3)
- Obtain weight
- Obtain vital signs (refer to Section 6.8.4)
- Assess presence and severity of ascites and hepatic encephalopathy for CPT score (refer to Section 6.8.7)
- Conduct pregnancy prevention counseling (only for females of childbearing potential and males with female partners of childbearing potential in the treatment group receiving RBV)
- Obtain blood samples for tests (approximately 35 mL of blood will be drawn total):
  - Hematology
  - Chemistry
  - Coagulation Tests
  - HCV RNA
  - Viral RNA Sequencing / Phenotyping Sample
  - HBV DNA Sample
- Obtain urine sample for:

— Pregnancy test for females of childbearing potential in the treatment group receiving RBV only (refer to Section 6.8.12)

## 6.5.3. Posttreatment Week 24 ( $\pm$ 5 days)

The following procedures/assessments are to be completed for all subjects, 24 weeks after taking the last dose of study drug:

- Perform complete physical examination (refer to Section 6.8.3)
- Obtain weight
- Obtain vital signs (refer to Section 6.8.4)
- Assess presence and severity of ascites and hepatic encephalopathy for CPT score (refer to Section 6.8.7)
- Obtain blood samples for tests (approximately 35 mL of blood will be drawn total):
  - Hematology
  - Chemistry
  - Coagulation Tests
  - HCV RNA
  - Viral RNA Sequencing / Phenotyping Sample
  - HBV DNA Sample
- Obtain urine sample for:
  - Pregnancy test for females of childbearing potential in the treatment group receiving RBV only (refer to Section 6.8.12)

#### 6.6. Early Termination (ET)

For subjects who have completed an ET visit, the posttreatment Week 4, 12, and 24 follow-up visits will be scheduled after the last dose of the study drugs.

When medically feasible, the medical monitor must be consulted prior to subject discontinuation.

The following procedures/assessments are to be completed at an Early Termination visit:

- Subject completes Health Related Quality of Life (HRQoL) surveys (refer to Section 6.8.6)
- Perform complete physical examination (refer to Section 6.8.3)

- Obtain weight
- Obtain vital signs (refer to Section 6.8.4)
- Assessment of AEs and concomitant medications
- Assess presence and severity of ascites and hepatic encephalopathy for CPT score (refer to Section 6.8.7)
- Conduct pregnancy prevention counseling
- Assess adherence with study drug dosing regimen including pill count. Collect any remaining study drug from the subject
- Obtain blood samples for tests (approximately 40 mL of blood will be drawn for required tests):
  - Hematology
  - Chemistry
  - Coagulation tests
  - HCV RNA
  - Viral RNA Sequencing / Phenotyping Sample
  - HBV DNA Sample
  - Single PK sample
  - Archive plasma sample (for subjects who have consented) (an additional 12 mL of blood will be drawn)
- Obtain urine sample for:
  - Pregnancy test for females of childbearing potential only

#### 6.7. Unscheduled Visit

A subject should attend an unscheduled visit if requested by the sponsor or the investigator. The assessments are at the investigator's discretion as clinically indicated, but the investigator should, at a minimum, collect AE and concomitant medication information. At all unscheduled visits initiated for the purpose of confirming virologic failure, a sample for a viral RNA sequencing/phenotyping must be collected.

## 6.8. Procedures and Specifications

#### **6.8.1.** Clinical Laboratory Analytes

<u>Hematology:</u> Hematocrit, Hemoglobin (Hb), Platelet count, Red blood cell count (RBC), White blood cell count (WBC) with differential (absolute and percentage) including Lymphocytes, Monocytes, Neutrophils, Eosinophils, and Basophils, Reticulocyte count and mean corpuscular volume (MCV).

<u>Coagulation:</u> INR, Prothrombin Activation %, Prothrombin time (PT), Activated partial thromboplastin time (aPTT)

<u>Chemistry:</u> Alanine aminotransferase (ALT/SGPT), Aspartate aminotransferase (AST/SGOT), Albumin, Alkaline phosphatase, Creatine Kinase, Creatinine, Direct Bilirubin, Total Bilirubin, Glucose, Lipase, Potassium, Sodium, phosphate, uric acid, FibroTest<sup>®</sup> (at Screening only).

<u>Urinalysis:</u> Blood, Glucose, Leukocyte esterase, pH, Protein, Urobilinogen. Reflex to microscopic urinalysis if dipstick result is abnormal.

<u>Virological Tests</u>: Serologies for HCV and HBV. HBV DNA (reflex testing done when ALT > 2x Day 1 value in subjects who are HBsAb or HBcAb positive at Screening). Serology and/or antigen testing for HIV, including reflex testing as necessary. HCV RNA will be measured using the COBAS<sup>®</sup> AmpliPrep/COBAS<sup>®</sup> TaqMan<sup>®</sup> HCV Quantitative Test, version 2.0. HCV genotype and subtype will be determined using the Siemens VERSANT<sup>®</sup> HCV Genotype INNO-LiPA2.0 Assay. Gilead reserves the right to use alternate assays for HCV RNA and HCV genotype should the above assays become unavailable or are not definitive.

IL28B genotype will be determined by polymerase chain reaction (PCR) amplification of the SNP, rs12979860, with sequence specific forward and reverse primers and allele specific fluorescently labeled TaqMan<sup>®</sup> MGB probes. Gilead reserves the rights to use an alternate assay for IL28B determination should the above assay become unavailable.

<u>Pregnancy Tests</u>: Serum β-hCG or Urine β-hCG (if positive, requires immediate confirmation with Serum β-hCG).

#### **6.8.2. Medical History**

Medical history, including details regarding illnesses and allergies, date(s) of onset, and whether condition(s) is currently ongoing, and medication history will be collected on all subjects during screening.

#### **6.8.3.** Complete Physical Examination

A physical examination must include source documentation of general appearance, and the following body systems: Head, neck, and thyroid; eyes, ears, nose, throat, mouth, and tongue; chest (excluding breasts); respiratory; cardiovascular; lymph nodes; abdomen; skin, hair, nails; musculoskeletal; neurological.

#### 6.8.4. Vital Signs

Assessment of vital signs will include measurement of resting blood pressure, pulse, respiratory rate, and temperature.

Blood pressure will be measured using the following standardized process:

- Subject should sit for  $\geq 5$  minutes with feet flat on the floor and measurement arm supported so that the midpoint of the manometer cuff is at heart level;
- Use a mercury sphygmomanometer or automatic blood pressure device with an appropriately sized cuff with the bladder centered over the brachial artery;
- Measure and record the blood pressure to the nearest 2 mmHg mark on the manometer or to the nearest whole number on an automatic device.

#### 6.8.5. 12-Lead ECG

Subjects will be required to rest in a supine position for  $\geq 5$  minutes prior to making a recording. The investigator (or qualified designee) should review the ECG traces recorded in real time for clinically significant abnormalities.

### 6.8.6. Health Related Quality of Life (HRQoL)

Health Related Quality of Life surveys (HRQoL) included in this study are the SF-36, Chronic Liver Disease Questionnaire (CLDQ-HCV), Fatigue Index (FACIT-F), and Work Productivity and Activity Impairment Questionnaire: Hepatitis C, v2.0 (WPAI: Hepatitis C).

The Health Related Quality of Life surveys (HRQoL) will only be administered to subjects if available at Day 1. The subject should read the questionnaire by himself/herself and record the answers by himself/herself.

#### **6.8.7. MELD and CPT Score Calculations**

MELD score and CPT score will be calculated from the central laboratory values attained at each visit. Assessment of ascites and hepatic encephalopathy will be determined by the site as in below table and will be entered into the eCRF. Besides calculating the CPT score at screening (using central laboratory values) and Day 1 (using local laboratory values) to determine eligibility, sites will not need to calculate these scores for subsequent visits.

#### 6.8.7.1. MELD Score

The MELD score is calculated using the following formula {MELD/PELD 2009}:

MELD = 3.8[serum bilirubin (mg/dL)] + 11.2[INR] + 9.57[serum creatinine\* (mg/dL)] + 6.43

Round to the nearest whole number. Laboratory values less than 1.0 are set to 1.0 for the purposes of the MELD score calculation.

#### 6.8.7.2. CPT Score

Child-Pugh-Turcotte score should be assessed at all visits per Table 6-1.

Table 6-1. Child-Pugh-Turcotte Classification of the severity of cirrhosis

| Measure | | 1 point | 2 points | 3 points |
|---|---|---|---|---|
| Total bilirubin, mg/dL, (μmol/L) | | <2, (<34) | 2-3, (34-50) | >3, (>50) |
| Serum albumin, g/dL | | >3.5 | 2.8-3.5 | <2.8 |
| Coagulation <sup>a</sup> | INR | < 1.7 | 1.7-2.3 | > 2.3 |
| | Prothrombin Activation % | >70% | 40-70% | <40% |
| Ascites <sup>b</sup> | | None No ascites and not on treatment for ascites | Mild/Moderate Cross sectional imaging showing ascites Abdominal distension Medication for ascites | Severe (diuretic-refractory) Visible clinically |
| Hepatic encephalopathy <sup>c</sup> | | None No encephalopathy and not on any treatment for hepatic encephalopathy | Medication-Controlled Subject is lethargic, may have moderate confusion Subject is receiving medical therapy for hepatic encephalopathy | Medication-Refractory Marked confusion/incoherent, rousable but sleeping unless aroused or comatosed |

a  $\;\;$  For coagulation, use either INR or Prothrombin activation %

- b {Moore et al 2003}
- c {Vilstrup et al 2014}

CPT <u>score</u> is obtained by adding the score for each parameter.

CPT <u>class</u>: A = 5-6 points

B = 7-9 points

C = 10-15 points

Records of concomitant medications for ascites and hepatic encephalopathy taken within 30 days of Screening through posttreatment Week 24 will be collected in the eCRF.

<sup>\*</sup> If subject has had dialysis twice within a week prior to the serum creatinine measurement, or is within 24 hours of continuous venovenous hemodiafiltration, then default to 4 mg/dL for serum creatinine value in MELD calculation.

#### **6.8.8.** Creatinine Clearance

Creatinine clearance is calculated by the Cockcroft-Gault equation {Cockcroft et al 1976} using actual body weight (ABW).

Male: 
$$CL_{cr} (mL/min) = [\underline{140 - age (years)}] \times ABW(kg)$$
  
 $72 \times S_{cr}$ 

Female: 
$$CL_{cr} (mL/min) = \underline{[140 - age (years)] \times ABW(kg) \times 0.85}$$
  
 $72 \times S_{cr}$ 

 $S_{cr}$  = serum creatinine (mg/dL)

For determination of eligibility, ideal body weight (IBW) may be used on a case-by-case basis when approved by the Medical Monitor.

## 6.8.9. Viral RNA Sequencing / Phenotyping Sample

Plasma samples will be collected at Day 1 and at on-treatment visits at Weeks 2, 4, 8, and 12 or early termination and all posttreatment visits and may be archived for viral sequence analysis. At any unscheduled visit initiated for the purpose of confirming virologic breakthrough, a viral sequence analysis plasma sample must be collected.

Details regarding the collection, processing, and shipping of samples will be included in the lab manual

#### 6.8.10. HBV DNA Sample

A sample for HBV DNA testing will be collected at on-treatment visits at Weeks 2, 4, 8, and 12 or early termination and all posttreatment visits. HBV DNA will only be tested when ALT > 2x Day 1 value in subjects who are HBsAb or HBcAb positive at Screening.

#### 6.8.11. Single Pharmacokinetic (PK) Sample

Single PK blood samples will be collected for all subjects at on-treatment visits at Weeks 2, 4, 8, and 12 or early termination and archived for PK analysis of SOF, its metabolites, VEL, and RBV (if appropriate). Approximately 6 mL of whole blood will be collected for each sample (which is included in the total blood volume amounts in Section 6.3). The exact time the study drugs were taken and whether or not the study drugs were taken with food on PK assessment days will be recorded in the source documents and eCRF.

Details regarding the collection, processing, and shipping of samples will be included in the lab manual.

## 6.8.12. Pregnancy Testing

All females of childbearing potential will have a serum pregnancy test at Screening. Urine pregnancy testing will occur at Day 1 and every 4 weeks through posttreatment 4.

Females of childbearing potential in the treatment group receiving RBV will have additional urine pregnancy testing every 4 weeks for a minimum of 6 months following last dose of RBV. If required by local regulations, additional pregnancy tests beyond 6 months may be added. In the event of a positive urine pregnancy result, subjects will be instructed to return to the clinic as soon as possible for a serum pregnancy test. Pregnancy test kits will be dispensed to female subjects of childbearing potential after the posttreatment Week 4 visit. The subject will be contacted by telephone monthly to confirm that urine pregnancy testing has been performed posttreatment and to record the outcome. Alternatively, if required by local regulations or preferred by the investigator or subject, the subject may return to the clinic for urine pregnancy tests.

#### 6.8.13. IL28B Testing

A blood sample will be obtained at Day 1 for specific genetic analysis of the rs12979860 (IL28B) genetic variant.

### 6.8.14. Archive Plasma Sample

For subjects who provide consent, an archive plasma sample (non-genetic) will be collected at Day 1 and Week 12 or ET (if applicable) visits. Approximately 12 mL of whole blood will be collected for each sample. The specimens collected will be used to increase our knowledge and understanding of the biology pathogenesis, progression and/or treatment outcomes, including efficacy, AEs, and the processes of drug absorption and disposition. These specimens may be used for retesting of the amount of HCV in the blood, clinical laboratory testing to provide additional clinical data and to develop non-genetic biomarker or diagnostic assays and establish the performance characteristics of these assays.

Details regarding the collection, processing, and shipping of samples will be included in the lab manual. At the conclusion of this study, these samples may be retained in storage by Gilead Sciences, Inc. for a period up to 15 years after the end of the study. These samples will be destroyed by internationally accepted means (eg, incineration).

#### 6.8.15. Genomic Testing






## 6.9. End of Study

Subjects are considered to have completed the study after the posttreatment Week 24 visit, regardless of treatment duration or early termination of study drugs.

# 6.10. Post Study Care

No poststudy ongoing care will be provided.

#### 7. ADVERSE EVENTS AND TOXICITY MANAGEMENT

# 7.1. Definitions of Adverse Events, Adverse Reactions, and Serious Adverse Events

#### 7.1.1. Adverse Events

An adverse event (AE) is any untoward medical occurrence in a clinical study subject administered a medicinal product, which does not necessarily have a causal relationship with the treatment. An AE can therefore be any unfavorable and/or unintended sign, symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs may also include pre- or posttreatment complications that occur as a result of protocol specified procedures, lack of efficacy, overdose, drug abuse/misuse reports, or occupational exposure. Preexisting events that increase in severity or change in nature during or as a consequence of participation in the clinical study will also be considered AEs.

An AE does not include the following:

- Medical or surgical procedures such as surgery, endoscopy, tooth extraction, and transfusion. The condition that led to the procedure may be an adverse event and must be reported.
- Pre-existing diseases, conditions, or laboratory abnormalities present or detected before the screening visit that do not worsen
- Situations where an untoward medical occurrence has not occurred (e.g., hospitalization for elective surgery, social and/or convenience admissions)
- Overdose without clinical sequelae (see Section 7.6.1)
- Any medical condition or clinically significant laboratory abnormality with an onset date before the consent form is signed and not related to a protocol-associated procedure is not an AE. It is considered to be pre-existing and should be documented on the medical history eCRF.

#### 7.1.2. Serious Adverse Events

A **serious adverse event** (SAE) is defined as an event that, at any dose, results in the following:

- Death
- Life-threatening (Note: The term "life-threatening" in the definition of "serious" refers to an event in which the subject was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if it were more severe.)
- In-patient hospitalization or prolongation of existing hospitalization

- Persistent or significant disability/incapacity
- A congenital anomaly/birth defect
- A medically important event or reaction: such events may not be immediately life-threatening or result in death or hospitalization but may jeopardize the subject or may require intervention to prevent one of the other outcomes constituting SAEs. Medical and scientific judgment must be exercised to determine whether such an event is a reportable under expedited reporting rules. Examples of medically important events include intensive treatment in an emergency room or at home for allergic bronchospasm; blood dyscrasias or convulsions that do not result in hospitalization; and development of drug dependency or drug abuse. For the avoidance of doubt, infections resulting from contaminated medicinal product will be considered a medically important event and subject to expedited reporting requirements.

# 7.1.3. Clinical Laboratory Abnormalities and Other Abnormal Assessments as Adverse Events or Serious Adverse Events

Laboratory abnormalities without clinical significance are not recorded as AEs or SAEs. However, laboratory abnormalities (eg, clinical chemistry, hematology, and urinalysis) that require medical or surgical intervention or lead to IMP interruption, modification, or discontinuation must be recorded as an AE, as well as an SAE, if applicable. In addition, laboratory or other abnormal assessments (eg, electrocardiogram, x-rays, vital signs) that are associated with signs and/or symptoms must be recorded as an AE or SAE if they meet the definition of an AE or SAE as described in Sections 7.1.1 and 7.1.2. If the laboratory abnormality is part of a syndrome, record the syndrome or diagnosis (eg, anemia), not the laboratory result (ie, decreased hemoglobin).

#### 7.2. Assessment of Adverse Events and Serious Adverse Events

The investigator or qualified subinvestigator is responsible for assessing AEs and SAEs for causality and severity, and for final review and confirmation of accuracy of event information and assessments.

## 7.2.1. Assessment of Causality for Study Drugs and Procedures

The investigator or qualified subinvestigator is responsible for assessing the relationship to study drug(s) therapy using clinical judgment and the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the IMP. For SAEs, an alternative causality must be provided (eg, pre-existing condition, underlying disease, intercurrent illness, or concomitant medication).
- Yes: There is reasonable possibility that the event may have been caused by the study drug(s).


It should be emphasized that ineffective treatment should not be considered as causally related in the context of adverse event reporting.

The relationship to study procedures (eg, invasive procedures such as venipuncture or biopsy) should be assessed using the following considerations:

- No: Evidence exists that the adverse event has an etiology other than the study procedure.
- Yes: The adverse event occurred as a result of protocol procedures, (eg, venipuncture)

## 7.2.2. Assessment of Severity

The severity grading of AEs will be assessed as Grade 1, 2, 3, or 4 using the GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities (Appendix 3). For AEs associated with laboratory abnormalities, the event should be graded on the basis of the clinical severity in the context of the underlying conditions; this may or may not be in agreement with the grading of the laboratory abnormality.

# 7.3. Investigator Requirements and Instructions for Reporting Adverse Events and Serious Adverse Events to Gilead or CRO

Requirements for collection prior to study drug(s) initiation:

After informed consent, but prior to initiation of study drug(s), the following types of events should be reported on the case report form (eCRF): all SAEs, and adverse events related to protocol-mandated procedures.

#### Adverse Events

Following initiation of study drug(s), collect all AEs, regardless of cause or relationship, until 30 days after last administration of study and report to the eCRF database as instructed.

All AEs should be followed up until resolution or until the adverse event is stable, if possible. Gilead Sciences may request that certain AEs be followed beyond the protocol defined follow up period.

#### Serious Adverse Events

All SAEs, regardless of cause or relationship, that occurs after the subject first consents to participate in the study (ie, signing the informed consent) and throughout the duration of the study, including the protocol-required post treatment follow-up period, must be reported to the eCRF database and Gilead Drug Safety and Public Health (DSPH) as instructed. This also includes any SAEs resulting from protocol-associated procedures performed after informed consent is signed.

Investigators are not obligated to actively seek SAEs after the protocol defined follow up period; however, if the investigator learns of any SAEs that occur after study participation has concluded

and the event is deemed relevant to the use of study drugs, he/she should promptly document and report the event to Gilead DSPH.

Prior treatment history is collected as part of the study entry criteria and evaluation of individual patient characteristics and will not be generating lack of effect reports as this is outside the scope of the present clinical study. However, investigators should report any cases of lack of effect that they feel appropriate regarding the previous treatment regimen as spontaneous reports to the relevant authorities or marketing authorisation holders.

• All AEs and SAEs will be recorded in the eCRF database within the timelines outlined in the eCRF completion guideline.

## Electronic Serious Adverse Event (eSAE) Reporting Process

- Site personnel record all SAE data in the eCRF database and from there transmit the SAE information to Gilead DSPH within 24 hours of the investigator's knowledge of the event. Detailed instructions can be found in the eCRF completion guidelines.
- If for any reason it is not possible to record the SAE information electronically, ie, the eCRF database is not functioning, record the SAE on the paper serious adverse event reporting form and submit within 24 hours as described above.

Fax: +1 (650) 522-5477

Gilead DSPH: Email: Safety FC@gilead.com

- As soon as it is possible to do so, any SAE reported via paper must be transcribed into the eCRF Database according to instructions in the eCRF completion guidelines.
- If an SAE has been reported via a paper form because the eCRF database has been locked, no further action is necessary.
- For fatal or life-threatening events, copies of hospital case reports, autopsy reports, and other
  documents are also to be submitted by e-mail or fax when requested and applicable.
   Transmission of such documents should occur without personal subject identification,
  maintaining the traceability of a document to the subject identifiers.
- Additional information may be requested to ensure the timely completion of accurate safety reports.
- Any medications necessary for treatment of the SAE must be recorded onto the concomitant medication section of the subject's eCRF and the event description section of the SAE form.

## 7.4. Gilead Reporting Requirements

Depending on relevant local legislation or regulations, including the applicable US FDA Code of Federal Regulations, the EU Clinical Trials Directive (2001/20/EC) and relevant updates, and other country-specific legislation or regulations, Gilead may be required to expedite to worldwide regulatory agencies reports of SAEs, serious adverse drug reactions (SADRs), or suspected unexpected serious adverse reactions (SUSARs). In accordance with the EU Clinical Trials Directive (2001/20/EC), Gilead or a specified designee will notify worldwide regulatory agencies and the relevant IEC in concerned Member States of applicable SUSARs as outlined in current regulations.

Assessment of expectedness for SAEs will be determined by Gilead using reference safety information specified in the investigator's brochure or relevant local label as applicable.

All investigators will receive a safety letter notifying them of relevant SUSAR reports associated with any study drug(s). The investigator should notify the IRB or IEC of SUSAR reports as soon as is practical, where this is required by local regulatory agencies, and in accordance with the local institutional policy.

## 7.5. Toxicity Management

### 7.5.1. RBV Dose Adjustments

Dose reduction or discontinuation of RBV due to toxicity is allowed at the discretion of the investigator. Once discontinued or reduced, the RBV dosing may be restarted or increased to the starting dose at the discretion of the investigator. RBV may be permanently discontinued due to toxicity without stopping SOF/VEL. Information on RBV dose reduction is provided in Table 7-1.

In the event a female partner of a male subject becomes pregnant, the male subject must permanently discontinue RBV, however they can continue SOF/VEL FDC.

Table 7-1. RBV Dose Reduction Recommendations

| Test items | Value | Ribavirin |
|---|---|---|
| Neutrophil count | < 500 /mm <sup>3</sup> | Discontinue |
| Platelet count | <50,000/mm <sup>3</sup> | Discontinue |
| | <25,000/mm <sup>3</sup> | Discontinue (resumption of dosing not allowed) |
| Hemoglobin level<br>(No cardiac disease or history of | < 11 g/dL at Week 1 to 4 after start<br>of administration | Reduce dose<br>600 mg/day → 200 mg/day |
| cardiac disease) | < 10 g/dL at Week 5 to 12 after<br>start of administration | $800 \text{ mg/day} \rightarrow 400 \text{ mg/day}$<br>$1,000 \text{ mg/day} \rightarrow 400 \text{ mg/day}$ |
| | < 8.5 g/dL | Discontinue |
| Hemoglobin level<br>(Cardiac disease or history of<br>cardiac disease present) | < 11 g/dL at Week 1 to 4 after start<br>of administration or during<br>administration, reduction of 2 g/dL<br>or more relative to Day 1 persists<br>for 4 weeks | uring $600 \text{ mg/day} \rightarrow 200 \text{ mg/day}$<br>of 2 g/dL $800 \text{ mg/day} \rightarrow 400 \text{ mg/day}$ |
| | < 10 g/dL at Week 5 to 12 after<br>start of administration or during<br>administration, reduction of 2 g/dL<br>or more relative to baseline persists<br>for 4 weeks | |
| | < 8.5 g/dL, or after dose reduction,<br>less than 12 g/dL even after 4<br>weeks | Discontinue |

Once RBV has been withheld due to either a laboratory abnormality or clinical manifestation, an attempt may be made to restart RBV at a lower daily dose with subsequent step-wise increase in the daily dose as clinically indicated. However, it is not recommended that the RBV daily dose be increased to the original assigned dose.

Subjects that require discontinuation of RBV for RBV-related events should continue with SOF/VEL for the remainder of the treatment period and complete all scheduled study visits.

#### 7.6. Special Situations Reports

## 7.6.1. Definitions of Special Situations

Special situation reports include all reports of medication error, abuse, misuse, overdose, reports of adverse events associated with product complaints, and pregnancy reports regardless of an associated AE.

Medication error is any unintentional error in the prescribing, dispensing, or administration of a medicinal product while in the control of the health care provider, subject, or consumer.

Abuse is defined as persistent or sporadic intentional excessive use of a medicinal product by a subject.

Misuse is defined as any intentional and inappropriate use of a medicinal product that is not in accordance with the protocol instructions or the local prescribing information.

An overdose is defined as an accidental or intentional administration of a quantity of a medicinal product given per administration or cumulatively which is above the maximum recommended dose as per protocol or in the product labelling (as it applies to the daily dose of the subject in question). In cases of a discrepancy in drug accountability, overdose will be established only when it is clear that the subject has taken the excess dose(s). Overdose cannot be established when the subject cannot account for the discrepancy except in cases in which the investigator has reason to suspect that the subject has taken the additional dose(s).

Product complaint is defined as complaints arising from potential deviations in the manufacture, packaging, or distribution of the medicinal product.

## 7.6.2. Instructions for Reporting Special Situations

## 7.6.2.1. Instructions for Reporting Pregnancies

The investigator should report pregnancies in female study subjects that are identified after initiation of study drug(s) and throughout the study, including the post study drug(s) follow-up period, to Gilead DSPH by transmitting electronically and also by sending paper pregnancy report form within 24 hours of becoming aware of the pregnancy.

Refer to Section 7.3 and the eCRF completion guidelines for full instructions on the mechanism of pregnancy reporting.

The pregnancy itself is not considered an AE nor is an induced elective abortion to terminate a pregnancy without medical reasons.

Any premature termination of pregnancy (eg, a spontaneous abortion, an induced therapeutic abortion due to complications or other medical reasons) must be reported within 24 hours as an SAE. The underlying medical reason for this procedure should be recorded as the AE term.

A spontaneous abortion is always considered to be an SAE and will be reported as described in Section 7.1.2. Furthermore, any SAE occurring as an adverse pregnancy outcome post study must be reported to Gilead DSPH.

The subject should receive appropriate monitoring and care until the conclusion of the pregnancy. The outcome should be reported to .Gilead DSPH using the pregnancy outcome report form. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead DSPH. Gilead DSPH contact information is as follows: Email: Safety FC@gilead.com and Fax: +1 (650) 522-5477.

Pregnancies of female partners of male study subjects exposed to other study drugs must also be reported and relevant information should be submitted to Gilead DSPH using the pregnancy and pregnancy outcome forms within 24 hours. Monitoring of the subject should continue until the conclusion of the pregnancy. If the end of the pregnancy occurs after the study has been completed, the outcome should be reported directly to Gilead DSPH, fax number +1 650 522-5477 or email Safety FC@gilead.com.

Clinical staff should also report any pregnancies to the Pregnancy Registry at 1 800-593-2214 (see also http://www.ribavirinpregnancyregistry.com). Refer to Appendix 4 for Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements.

## 7.6.2.2. Reporting Other Special Situations

All other special situation reports must be reported on electronic special situations report form and transmitted to Gilead DSPH within 24 hours of the investigator becoming aware of the situation. If for any reason it is not possible to record the special situation report (SSR) information electronically, ie, the eCRF database is not functioning, record the SSR on the paper special situation reporting form and submit within 24 hours to:

Gilead DSPH: Fax: +1 (650) 522-5477

Email: Safety\_FC@gilead.com

As soon as it is possible to do so, any SSR reported via paper must be transcribed into the eCRF Database according to instructions in the eCRF completion guidelines.

These reports must consist of situations that involve study drug(s) and/or Gilead concomitant medications, but do not apply to non-Gilead concomitant medications.

Special situations involving non-Gilead concomitant medications does not need to be reported on the special situations report form; however, for special situations that result in AEs due to a non-Gilead concomitant medication, the AE should be reported on the AE form.

Any inappropriate use of concomitant medications prohibited by this protocol should not be reported as "misuse," but may be more appropriately documented as a protocol deviation.

Refer to Section 7.3 and the eCRF completion guidelines for full instructions on the mechanism of special situations reporting.

All clinical sequelae in relation to these special situation reports will be reported as AEs or SAEs at the same time using the AE eCRF and/or the SAE report form. Details of the symptoms and signs, clinical management, and outcome will be reported, when available.

#### 8. STATISTICAL CONSIDERATIONS

## 8.1. Analysis Objectives and Endpoints

#### 8.1.1. Analysis Objectives

The primary objectives of this study are:

- To evaluate the antiviral efficacy of therapy with sofosbuvir/velpatasvir (SOF/VEL)
  fixed-dose combination (FDC) with or without ribavirin for 12 weeks as measured by the
  proportion of subjects with sustained virologic response 12 weeks after cessation of treatment
  (SVR12)
- To evaluate the safety and tolerability of each treatment regimen

The secondary objectives of this study are:

- To determine the proportion of subjects who attain SVR at 4 and 24 weeks after cessation of treatment (SVR4 and SVR24)
- To evaluate the proportion of subjects with virologic failure
- To evaluate the rapeutic efficacy as measured by the change of CPT score and MELD score
- To evaluate the kinetics of circulating HCV RNA during treatment and after cessation of treatment
- To evaluate the emergence of viral resistance to SOF and VEL during treatment and after cessation of treatment

The exploratory objectives of this study are:



#### 8.1.2. Primary Endpoint

The primary efficacy endpoint is SVR12 (HCV RNA < LLOQ 12 weeks after cessation of treatment) in the Full Analysis Set (FAS) population.

The primary safety endpoint is any AE leading to permanent discontinuation of study drugs.

## 8.1.3. Secondary Endpoint

The secondary efficacy endpoints include the following:

- The proportion of subjects with HCV RNA < LLOQ at 4 and 24 weeks after cessation of treatment (SVR4 and SVR24)
- Proportion of subjects who have HCV RNA < LLOQ by visit while on treatment
- MELD and CPT score changes from Baseline
- HCV RNA change from Baseline
- The proportion of subjects with virologic failure

## 8.1.4. Other Endpoints of Interest

Additional efficacy evaluations may include the health related quality of life endpoints.

## 8.2. Analysis Conventions

All individual subject data will be listed as measured. All statistical summaries and analyses will be performed using SAS® software (SAS Institute, Cary, North Carolina, USA).

The study drugs in this study include SOF/VEL FDC and RBV. Last dose of study drugs refers to the last dose of the study drugs in a treatment group and will be used in the definition of treatment-emergent AEs and laboratory abnormalities as well as the efficacy endpoints of SVR at various post treatment time points.

#### 8.2.1. Analysis Sets

#### 8.2.1.1. Efficacy

The primary analysis set for efficacy analysis is defined as the Full Analysis Set (FAS) which includes all randomized subjects who took at least 1 dose of study drug(s).

## 8.2.1.2. Safety

The primary analysis set for safety analyses will include all subjects who took at least 1 dose of study drug(s). Treatment-emergent data will be analyzed and defined as data collected from the first dose of study drugs through the date of last dose of study drugs plus 30 days.

#### 8.2.1.3. Pharmacokinetics

The Pharmacokinetic (PK) Analysis Set includes all subjects who took at least 1 dose of the study drugs and have at least 1 nonmissing concentration value for the corresponding analyte in

plasma. The analyte of interest may include SOF, GS-566500, GS-331007, VEL, and RBV (if appropriate). The PK analysis set will be used for analyses of general PK.

## 8.3. Data Handling Conventions

Missing data can have an impact upon the interpretation of the trial data. Other than the endpoints discussed below, values for missing data will not be imputed.

For the analyses of categorical HCV RNA data, missing posttreatment HCV RNA data will have the missing data imputed. Missing on-treatment HCV RNA will have the missing data imputed up to the time of the last dose.

If a data point is missing and is preceded and followed in time by values that are "< LLOQ target not detected (TND)," then the missing data point will be set to "< LLOQ TND." If a data point is missing and preceded and followed by values that are "< LLOQ detected," or preceded by "< LLOQ detected" and followed by "< LLOQ TND," or preceded by "< LLOQ TND" and followed by "< LLOQ detected," then the missing value will be set to "< LLOQ detected." In these situations the data point will be termed a bracketed success; otherwise, the data point will be termed a bracketed failure (i.e.,  $\geq$  LLOQ detected). If a data point is missing and is not bracketed, the missing data point will also be termed a failure (i.e.,  $\geq$  LLOQ detected) except for SVR24, which will be imputed according to the SVR12 status. Success for SVR12 who have no further HCV RNA measurements collected will be counted as a success for SVR24 due to the high correlation between these 2 endpoints.

Where appropriate, safety data for subjects that did not complete the study will be included in summary statistics. For example,

- If a subject took at least 1 dose of study drugs, the subject will be included in a summary of AEs according to the treatment received; otherwise, if the subject is not dosed, then they will be excluded from the summary.
- If safety laboratory results for a subject are missing for any reason at a time point, the subject will be excluded from the calculation of summary statistics for that time point. If the subject is missing a pre-dose value, then the subject will be excluded from the calculation of summary statistics for the pre-dose value and the change from pre-dose values.

Values for missing safety laboratory data will not be imputed; however, a missing baseline result will be replaced with a screening result, if available. If no pre-treatment safety laboratory value is available, the baseline value will be assumed to be normal (ie, no grade [Grade 0]) in the summary of graded laboratory abnormalities. Values for missing vital signs data will not be imputed; however, a missing baseline result will be replaced with a screening result, if available.

HCV RNA values below the LLOQ for the assay will be set to the lower limit minus 1 for calculation of summary statistics for the actual HCV RNA values and the change from baseline values by study visit. The reported values will be provided in the HCV RNA listing.

For selected analyses of early time point data, HCV RNA data (IU/mL) may be transformed to the logarithmic (base 10) scale (log<sub>10</sub> IU/mL).

For PK plasma/blood concentrations and analysis of PK parameters natural logarithmic transformation will be used.

#### 8.4. Demographic Data and Baseline Characteristics

Demographic and baseline measurements will be summarized using standard descriptive methods.

Demographic data will include age, sex, self-identified race and ethnicity. Baseline characteristic data will include body mass index, HCV RNA level (log<sub>10</sub> IU/mL), genotype of HCV infection, IL28B genotype, CPT, MELD scores and additional endpoints as necessary.

## 8.5. Efficacy Analysis

## 8.5.1. Primary Analysis

The primary efficacy endpoint for this study will be the proportion of subjects with SVR12, defined as HCV RNA < LLOQ 12 weeks after cessation of treatment. The primary analysis will be performed after all randomized and treated subjects have been followed through 12 weeks posttreatment or discontinued from study.

A point estimate with a two-sided 95% exact confidence interval using the binomial distribution (Clopper-Pearson method) will be constructed for the SVR12 rate by treatment group.

In the primary efficacy analysis, the SVR12 rate in each of the 2 treatment groups will be compared to the spontaneous clearance rate of 1% using two-sided exact one-sample binomial test with Bonferroni alpha adjustment (each at significance level 0.025): ie, for each treatment group the hypothesis for superiority is as follows:

H0: SVR12 rate = 1%, H1: SVR12 rate  $\neq 1\%$ 

This 1% spontaneous rate was assumed in the statistical test of treatment benefit because there are no currently available treatment options for these subjects and non-treatment rarely results in spontaneous cure.

#### 8.5.2. Secondary Analyses

The proportion of subjects with HCV RNA below LLOQ over time (including SVR endpoints) will be presented in tabular and graphical form.

Descriptive summaries and listings will be provided for additional efficacy evaluations including HCV RNA values and change from baseline through end of treatment, MELD and CPT scores and change from Baseline, and subjects who experience virologic failure.



Details on efficacy analyses will be described in the statistical analysis plan.

#### 8.6. Safety Analysis

Safety will be evaluated by assessment of clinical laboratory tests, physical examinations, and vital signs measurements and AEs will be documented at various time points during the study.

All safety data collected, on or after the first dose of study drugs administration up to 30 days after the last dose of study drugs will be summarized by treatment group according to the study drugs received.

#### 8.6.1. Extent of Exposure

A subject's extent of exposure to the study drug will be generated from the study drug administration page of eCRF. Exposure data will be summarized by treatment group.

#### 8.6.2. Adverse Events

Clinical and laboratory adverse events will be coded using the Medical Dictionary for Regulatory Activities (MedDRA). System Organ Class (SOC), High-Level Group Term (HLGT), High-Level Term (HLT), Preferred Term (PT), and Lower-Level Term (LLT) will be attached to the clinical database.

Events will be summarized on the basis of the date of onset for the event. A treatment-emergent adverse event will be defined as any AE with an onset date on or after the study drugs start date and no later than 30 days after permanent discontinuation of the study drugs; or any AE leading to premature discontinuation of the study drugs.

Summaries (number and percentage of subjects) or listings, as appropriate, of treatmentemergent adverse events (by SOC, and PT) will be provided by treatment group for:

- All AEs
- AEs of Grade 3 or above
- AEs of Grade 2 or above
- All treatment-related AEs.
- Treatment-related AEs of Grade 3 or above
- Treatment-related AEs of Grade 2 or above

- All SAEs
- All treatment-related SAEs
- AEs leading to premature discontinuation of any study drugs
- AEs leading to modification or interruption of any study drugs

All AEs collected during the course of the study will be presented in data listings.

## 8.6.3. Laboratory Evaluations

Selected laboratory data will be summarized (n, mean, SD, median, Q1, Q3, minimum, and maximum) by treatment group and study visit along with corresponding change from baseline.

Graded laboratory abnormalities will be defined using the laboratory toxicity grading scheme defined in Appendix 3 of this protocol. The incidence of treatment emergent laboratory abnormalities, defined as values that increase by at least one toxicity grade from baseline at any time post-baseline up to the date of last dose of study drugs plus 30 days will be summarized.

Values for missing safety laboratory data will not be imputed; however, a missing Day 1 result will be replaced with a screening result, if available. If no pretreatment laboratory value is available, the Day 1 value will be assumed to be normal (i.e., no grade [Grade 0]) for the summary of graded laboratory abnormalities. If Day 1 data are missing, then any post-baseline graded abnormality (ie, at least Grade 1) will be considered treatment emergent.

All laboratory abnormalities will be included in the listings of laboratory data.

#### 8.6.4. Other Safety Evaluations

Individual data for vital signs measurements will be listed by subject and summarized by treatment group by descriptive statistical summaries (n, mean, SD, median, Q1, Q3, minimum, and maximum), as appropriate.

## 8.7. Pharmacokinetic Analysis

In the PK analysis set, concentrations of SOF, its metabolites GS-566500 and GS-331007, VEL, and RBV (if appropriate) in plasma may be determined using validated bioanalytical assays and listed. Details of the analyses will be provided in the pharmacokinetic reporting and analysis plan.

#### 8.8. Sample Size

A sample size of 50 subjects in each treatment group will provide over 99% power to detect at least 40% improvement in SVR12 rate from the assumed spontaneous rate of 1% or less using a two-sided exact one-sample binomial test at significance level of 0.025.

## 8.9. Data Monitoring Committee

An external multidisciplinary data monitoring committee (DMC) will perform a review of accumulated safety data from the first 20 subjects with CPT B cirrhosis at Screening enrolled through 4 weeks of treatment (or treatment discontinuation) and provide a recommendation to Gilead on whether these data support enrollment of subjects with CPT C cirrhosis at Screening. The DMC may also provide recommendations as needed regarding study design, conduct, and the need for additional meetings.

The DMC's specific activities will be defined by a mutually agreed charter, which will define the DMC's membership, conduct and meeting schedule.

While the DMC will be asked to advise Gilead regarding future conduct of the study, including possible early study termination, Gilead retains final decision-making authority on all aspects of the study.

#### 9. **RESPONSIBILITIES**

## 9.1. Investigator Responsibilities

#### 9.1.1. Good Clinical Practice

The investigator will ensure that this study is conducted in accordance with the principles of the Declaration of Helsinki (as amended in Edinburgh, Tokyo, Venice, Hong Kong, and South Africa), International Conference on Harmonisation (ICH) guidelines, or with the laws and regulations of the country in which the research is conducted, whichever affords the greater protection to the study subject.

This protocol is to be conducted in accordance with the guidance stipulated in Article 14, Paragraph 3 and Article 80-2 of the Law for Ensuring the Quality, Efficacy, and Safety of Drugs and Medical Devices, "MHLW Ordinance on Good Clinical Practice" {Ministry of Health and Welfare 2013}.

The investigator and all applicable subinvestigators will comply with 21 CFR, Part 54, 1998, providing documentation of their financial interest or arrangements with Gilead, or proprietary interests in the investigational drug under study. This documentation must be provided prior to the investigator's (and any subinvestigator's) participation in the study. The investigator and subinvestigator agree to notify Gilead of any change in reportable interests during the study and for 1 year following completion of the study. Study completion is defined as the date when the last subject completes the protocol-defined activities.

# 9.1.2. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) Review and Approval

The investigator (or sponsor as appropriate according to local regulations) will submit this protocol, informed consent form, and any accompanying material to be provided to the subject (such as advertisements, subject information sheets, or descriptions of the study used to obtain informed consent) to an IRB or IEC. The investigator will not begin any study subject activities until approval from the IRB or IEC has been documented and provided as a letter to the investigator.

Before implementation, the investigator will submit to and receive documented approval from the IRB or IEC any modifications made to the protocol or any accompanying material to be provided to the subject after initial approval, with the exception of those necessary to reduce immediate risk to study subjects.

#### 9.1.3. Informed Consent

The investigator is responsible for obtaining written informed consent from each individual participating in this study after adequate explanation of the aims, methods, objectives, and potential hazards of the study and before undertaking any study-related procedures. The

investigator must use the most current approved consent form for documenting written informed consent. Each informed consent will be appropriately signed and dated by the subject and the person conducting the consent discussion, and also by an impartial witness if required by local requirements. The consent form will inform subjects about genomic testing and sample retention.

### 9.1.4. Confidentiality

The investigator must assure that subjects' anonymity will be strictly maintained and that their identities are protected from unauthorized parties. Only subject initials, date of birth, another unique identifier (as allowed by local law), and an identification code will be recorded on any form or biological sample submitted to the Sponsor, IRB or IEC, or laboratory. Laboratory specimens must be labeled in such a way as to protect subject identity while allowing the results to be recorded to the proper subject. Refer to specific laboratory instructions. NOTE: The investigator must keep a screening log showing codes, names, and addresses for all subjects screened and for all subjects enrolled in the trial. Subject data will be processed in accordance with all applicable regulations.

The investigator agrees that all information received from Gilead, including but not limited to the investigator brochure, this protocol, eCRF, the study drugs, and any other study information, remain the sole and exclusive property of Gilead during the conduct of the study and thereafter. This information is not to be disclosed to any third party (except employees or agents directly involved in the conduct of the study or as required by law) without prior written consent from Gilead. The investigator further agrees to take all reasonable precautions to prevent the disclosure by any employee or agent of the study site to any third party or otherwise into the public domain.

#### 9.1.5. Study Files and Retention of Records

The investigator must maintain adequate and accurate records to enable the conduct of the study to be fully documented and the study data to be subsequently verified. These documents should be classified into at least the following two categories: (1) investigator's study file, and (2) subject clinical source documents.

The investigator's study file will contain the protocol/amendments, and governmental approval with correspondence, informed consent, drug records, staff curriculum vitae and authorization forms, and other appropriate documents and correspondence.

The required source data should include sequential notes containing at least the following information for each subject:

- Subject identification (name, date of birth, gender);
- Documentation that subject meets eligibility criteria, ie, history, physical examination, and confirmation of diagnosis (to support inclusion and exclusion criteria);
- Documentation of the reason(s) a consented subject is not enrolled;


- Participation in study (including study number);
- Study discussed and date of informed consent;
- Dates of all visits;
- Documentation that protocol specific procedures were performed;
- Results of efficacy parameters, as required by the protocol;
- Start and end date (including dose regimen) of study drugs, including dates of dispensing and return;
- Record of all adverse events and other safety parameters (start and end date, and including causality and severity);
- Concomitant medication (including start and end date, dose if relevant; dose changes);
- Date of study completion and reason for early discontinuation, if it occurs.

All clinical study documents must be retained by the investigator until at least 2 years or according to local laws, whichever is longer, after the last approval of a marketing application in an ICH region (ie, United States, Europe, or Japan) and until there are no pending or planned marketing applications in an ICH region; or, if no application is filed or if the application is not approved for such indication, until 2 years after the investigation is discontinued and regulatory authorities have been notified. Investigators may be required to retain documents longer if specified by regulatory requirements, by local regulations, or by an agreement with Gilead. The investigator must notify Gilead before destroying any clinical study records.

Should the investigator wish to assign the study records to another party or move them to another location, Gilead must be notified in advance.

If the investigator cannot provide for this archiving requirement at the study site for any or all of the documents, special arrangements must be made between the investigator and Gilead to store these records securely away from the site so that they can be returned sealed to the investigator in case of an inspection. When source documents are required for the continued care of the subject, appropriate copies should be made for storage away from the site.

## 9.1.6. Case Report Forms

For each subject consented, an eCRF will be completed by an authorized study staff member whose training for this function is documented according to study procedures. eCRF should be completed on the day of the subject visit to enable the sponsor to perform central monitoring of safety data. The Eligibility Criteria eCRF should be completed only after all data related to eligibility have been received. Subsequent to data entry, a study monitor will perform source data verification within the EDC system. Original entries as well as any changes to data fields


will be stored in the audit trail of the system. Prior to database lock (or any interim time points as described in the clinical data management plan), the investigator will use his/her log-in credentials to confirm that the forms have been reviewed, and that the entries accurately reflect the information in the source documents. The eCRF capture the data required per the protocol schedule of events and procedures. System-generated or manual queries will be issued to the investigative site staff as data discrepancies are identified by the monitor or internal Gilead staff, who routinely review the data for completeness, correctness, and consistency. The site coordinator is responsible for responding to the queries in a timely manner, within the system, either by confirming the data as correct or updating the original entry, and providing the reason for the update (eg, data entry error). At the conclusion of the trial, Gilead will provide the site with a read-only archive copy of the data entered by that site. This archive must be stored in accordance with the records retention requirements outlined in Section 9.1.5.

#### 9.1.7. Study Drug Accountability and Return

Gilead recommends that used and unused study drugs supplies be returned to the shipping facility from which it came for eventual destruction. The study monitor will provide instructions for return. If return is not possible, the study monitor will evaluate each study center's study drugs disposal procedures and provide appropriate instruction for destruction of unused study drugs supplies. If the site has an appropriate standard operating procedure (SOP) for drug destruction as determined by Gilead, the site may destroy used (empty or partially empty) and unused study drugs supplies in accordance with that site's approved SOP. A copy of the site's approved SOP will be obtained for central files.

If study drugs are destroyed on site, the investigator or designee (ie, pharmacist) must maintain accurate records for all study drugs destroyed. Records must show the identification and quantity of each unit destroyed, the method of destruction, and the person who disposed of the study drugs. Upon study completion, originals of the study drugs accountability records must be filed at the site. A copy will be returned to Gilead.

The study monitor will review study drugs supplies and associated records at periodic intervals.

#### 9.1.8. Inspections

The investigator will make available all source documents and other records for this trial to Gilead's appointed study monitors, to IRB/IECs, or to regulatory authority or health authority inspectors.

### 9.1.9. Protocol Compliance

The investigator is responsible for ensuring the study is conducted in accordance with the procedures and evaluations described in this protocol.

## 9.2. Sponsor Responsibilities

#### 9.2.1. Protocol Modifications

Protocol modifications, except those intended to reduce immediate risk to study subjects, may be made only by Gilead. The investigator must submit all protocol modifications to the IRB or IEC in accordance with local requirements and receive documented approval before modifications can be implemented.

## 9.2.2. Study Report and Publications

A clinical study report (CSR) will be prepared and provided to the regulatory agency. Gilead will ensure that the report meets the standards set out in the ICH Guideline for Structure and Content of Clinical Study Reports (ICH E3). Note that an abbreviated report may be prepared in certain cases.

Investigators in this study may communicate, orally present, or publish in scientific journals or other scholarly media only after the following conditions have been met:

The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form or the study has been completed at all study sites for at least 2 years.

The investigator will submit to Gilead any proposed publication or presentation along with the respective scientific journal or presentation forum at least 30 days before submission of the publication or presentation.

No such communication, presentation, or publication will include Gilead's confidential information (see Section 9.1.4).

The investigator will comply with Gilead's request to delete references to its confidential information (other than the study results) in any paper or presentation and agrees to withhold publication or presentation for an additional 60 days in order to obtain patent protection if deemed necessary.

## 9.3. Joint Investigator/Sponsor Responsibilities

#### 9.3.1. Access to Information for Monitoring

In accordance with ICH Good Clinical Practice (ICH GCP) guidelines, the study monitor must have direct access to the investigator's source documentation in order to verify the accuracy of the data recorded in the eCRF.

The monitor is responsible for routine review of the eCRF at regular intervals throughout the study to verify adherence to the protocol and the completeness, consistency, and accuracy of the data being entered on them. The monitor should have access to any subject records needed to

verify the entries on the eCRF. The investigator agrees to cooperate with the monitor to ensure that any problems detected through any type of monitoring (central, on site) are resolved.

## 9.3.2. Access to Information for Auditing or Inspections

Representatives of regulatory authorities or of Gilead may conduct inspections or audits of the clinical study. If the investigator is notified of an inspection by a regulatory authority the investigator agrees to notify Gilead or the CRO immediately. The investigator agrees to provide to representatives of a regulatory agency or Gilead access to records, facilities, and personnel for the effective conduct of any inspection or audit.

## 9.3.3. Study Discontinuation

Both the sponsor and the investigator reserve the right to terminate the study at any time. Should this be necessary, both parties will arrange discontinuation procedures and notify the appropriate regulatory authority(ies), IRBs, and IECs. In terminating the study, Gilead and the investigator will assure that adequate consideration is given to the protection of the subjects' interests.
#### 10. REFERENCES

- Allison RD, Tong X, Moorman AC, Ly KN, Rupp L, Xu F, et al. Increased Incidence of Cancer and Cancer-related Mortality Among Persons with Chronic Hepatitis C Infection, 2006-2010. J Hepatol 2015.
- Arias A, Aguilera A, Soriano V, Benitez-Gutierrez L, Lledo G, Navarro D, et al. Rate and predictors of treatment failure to all-oral HCV regimens outside clinical trials. Antivir Ther 2016.
- Charlton M, Everson GT, Flamm SL, Kumar P, Landis C, Brown Jr RS, et al. Ledipasvir and Sofosbuvir Plus Ribavirin for Treatment of HCV Infection in Patients with Advanced Liver Disease. Gastroenterology 2015:649-59.
- Chung H, Ueda T, Kudo M. Changing trends in hepatitis C infection over the past 50 years in Japan. Intervirology 2010;53 (1):39-43.
- Cockcroft DW, Gault MH. Prediction of creatinine clearance from serum creatinine. Nephron 1976;16:31-41.
- Curry MP, O'Leary JG, Bzowej N, Muir AJ, Korenblat KM, Fenkel JM, et al. Sofosbuvir and Velpatasvir for HCV in Patients with Decompensated Cirrhosis. N Engl J Med 2015.
- Gilead Sciences Inc. SOVALDI® (sofosbuvir) tablets, for oral use. US Prescribing Information. Foster City, CA. December 2013:
- Gilead Sciences Inc. EPCLUSA® (sofosbuvir and velpatasvir) tablets, for oral use. US Prescribing Information. Foster City, CA. Revised June. 2016a:
- Gilead Sciences Inc. HARVONI® (ledipasvir and sofosbuvir) tablets, for oral use. U.S. Prescribing Information. Foster City, CA. Revised June. 2016b:
- Gilead Sciences International Ltd. Epclusa 400 mg/100 mg film-coated tablets (SmPC). 2016:41.
- Gilead Sciences International Ltd. HARVONI (ledipasvir/sofosbuvir) 90 mg/400 mg Film-Coated Tablets. Summary of Product Characteristics. Cambridge, UK. Revised April. 2016:
- Gower E, Estes C, Blach S, Razavi-Shearer K, Razavi H. Global epidemiology and genotype distribution of the hepatitis C virus infection. J Hepatol 2014.


- Ioannou GN, Beste LA, Chang MF, Green PK, Lowey E, Tsui JI, et al. Effectiveness of Sofosbuvir, Ledipasvir/Sofosbuvir, or Paritaprevir/Ritonavir/Ombitasvir and Dasabuvir Regimens for Treatment of Patients With Hepatitis C in the Veterans Affairs National Healthcare System [Accepted Manuscript]. Gastroenterology 2016.
- Manns M, Samuel D, Gane EJ, Mutimer D, McCaughan G, Buti M, et al. Ledipasvir and sofosbuvir plus ribavirin in patients with genotype 1 or 4 hepatitis C virus infection and advanced liver disease: a multicentre, open-label, randomised, phase 2 trial. Lancet Infect Dis 2016.
- MELD/PELD. Calculator Documentation. 28 January. 2009:
- Ministry of Health and Welfare. Ministerial Ordinance on Good Clinical Practice for Drugs. Ordinance of the Ministry of Health and Welfare No. 28 of March 27, 1997 (As last amended by the Ordinance of Ministry of Health, Labour and Welfare No. 161 of December 28, 2012). Provisional Translation as of March 2013.
- Moore KP, Wong F, Gines P, Bernardi M, Ochs A, Salerno F, et al. The management of ascites in cirrhosis: report on the consensus conference of the International Ascites Club. Hepatology 2003;38 (1):258-66.
- Morgan RL, Baack B, Smith BD, Yartel A, Pitasi M, Falck-Ytter Y. Eradication of Hepatitis C Virus Infection and the Development of Hepatocellular Carcinoma. Ann Intern Med 2013;158 (5 (Part I)).
- MSD K.K. Kudan-kita Chiyoda-ku. REBETOL® (ribavirin) Capsules 200 mg. Japan Prescribing Information [English]. Tokyo, Japan. Revised January. 2016:
- Perz JF, Armstrong GL, Farrington LA, Hutin YJ, Bell BP. The contributions of hepatitis B virus and hepatitis C virus infections to cirrhosis and primary liver cancer worldwide. J Hepatol 2006;45 (4):529-38.
- Poynard T, McHutchison J, Manns M, Trepo C, Lindsay K, Goodman Z, et al. Impact of pegylated interferon alfa-2b and ribavirin on liver fibrosis in patients with chronic hepatitis C. Gastroenterology 2002;122 (5):1303-13.
- Sievert W, Altraif I, Razavi HA, Abdo A, Ahmed EA, Alomair A, et al. A systematic review of hepatitis C virus epidemiology in Asia, Australia and Egypt. Liver Int 2011;31 Suppl 2:61-80.
- Tanaka J, Kumagai J, Katayama K, Komiya Y, Mizui M, Yamanaka R, et al. Sex- and agespecific carriers of hepatitis B and C viruses in Japan estimated by the prevalence in the 3,485,648 first-time blood donors during 1995-2000. Intervirology 2004;47 (1):32-40.


- Thein HH, Yi Q, Dore GJ, Krahn MD. Estimation of stage-specific fibrosis progression rates in chronic hepatitis C virus infection: a meta-analysis and meta-regression. Hepatology 2008;48 (2):418-31.
- van der Meer AJ, Veldt BJ, Feld JJ, Wedemeyer H, Dufour JF, Lammert F, et al. Association between sustained virological response and all-cause mortality among patients with chronic hepatitis C and advanced hepatic fibrosis. JAMA 2012;308 (24):2584-93.
- Veldt BJ, Heathcote EJ, Wedemeyer H, Reichen J, Hofmann WP, Zeuzem S, et al. Sustained virologic response and clinical outcomes in patients with chronic hepatitis C and advanced fibrosis. Ann Intern Med 2007;147 (10):677-84.
- Vilstrup H, Amodio P, Bajaj J, Cordoba J, Ferenci P, Mullen KD, et al. Hepatic encephalopathy in chronic liver disease: 2014 Practice Guideline by the American Association for the Study of Liver Diseases and the European Association for the Study of the Liver. Hepatology 2014;60 (2):715-35.
- World Health Organization (WHO). Media Centre: Hepatitis C Fact Sheet. Updated July. 2016.

# 11. APPENDICES

| Appendix 1. | Investigator Signature Page |
|-------------|-----------------------------|
| Appendix 2. | Study Procedures Table |

Appendix 3. GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities Appendix 4. Pregnancy Precautions, Definition for Female of Childbearing Potential, and

Contraceptive Requirements

#### Appendix 1. **Investigator Signature Page**

GILEAD SCIENCES, INC. 333 LAKESIDE DRIVE FOSTER CITY, CA 94404

## STUDY ACKNOWLEDGEMENT

| A Multicenter, Randomized, Phase 3, Open-Label<br>Sofosbuvir/Velpatasvir ± Ribavirin for 12 Week<br>Decompensate | s in Subjects with Chronic HCV Infection and |
|---|---|
| GS-US-342-4019, Protocol Ame | ndment 1, 17 November 2016 |
| This protocol has been approved by Gilead Science this approval. And Osinusi, MD, MPH (Printed) | PPD Signature |
| Nov 17, 2016 Date | |
| INVESTIGATOR | STATEMENT |
| I have read the protocol, including all appendices, details for me and my staff to conduct this study as outlined herein and will make a reasonable effort t designated. | s described. I will conduct this study as |
| I will provide all study personnel under my supervinformation provided by Gilead Sciences, Inc. I withat they are fully informed about the drugs and the | ill discuss this material with them to ensure |
| Principal Investigator Name (Printed) | Signature |
| Date | Site Number |

**Appendix 2. Study Procedures Table** 

| | | | | | | | | | tmen<br>±3 da | ıt We<br>ays) | ek | | | | | ttreatm<br>k (±5 c | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Day 1 <sup>a</sup> | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12/ET <sup>b</sup> | 4 | 12 | 24 |
| Clinical Assessments | | | | | | | | | | | | | | | | | |
| Informed Consent | X | | | | | | | | | | | | | | | | |
| Determine Eligibility | X | X | | | | | | | | | | | | | | | |
| Verification of CPT score <sup>c</sup> | | X | | | | | | | | | | | | | | | |
| Medical History | X | | | | | | | | | | | | | | | | |
| Physical Examination | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Height | X | | | | | | | | | | | | | | | | |
| Weight | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Vital Signs <sup>d</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 12-Lead ECG <sup>e</sup> | X | X | | | | | | | | | | | | | | | |
| Adverse Events and Concomitant<br>Medications <sup>f</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Pregnancy Prevention Counseling | | X | | | | X | | | | X | | | | X | X | X | |
| Health Related Quality of Life <sup>g</sup> | | X | | | | | | | | | | | | X | | X | |
| Assessment of ascites and hepatic encephalopathy | X | X | | | | X | | | | X | | | | X | X | X | X |
| Imaging for HCC <sup>h</sup> | X | | | | | | | | | | | | | | | | |
| Review of Study Drug Adherence and Drug<br>Accountability <sup>i</sup> | | | X | X | X | X | X | X | X | X | X | X | X | X | | | |
| Study Drug Dispensing <sup>j</sup> | | X | | | | X | | | | X | | | | | | | |
| Close Monitoring of Subjects with CPT C Cirrhosis <sup>k</sup> | | X | | | | | | | | | | | | | | | |

| | | Treatment Week Posttreatmen (±3 days) Week (±5 day | | | | | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | Screening | Day 1 <sup>a</sup> | 1 | 2 | 3 | 4 | 5 | 6 | 7 | 8 | 9 | 10 | 11 | 12/ET <sup>b</sup> | 4 | 12 | 24 |
| <b>Laboratory Assessments</b> | | | | | | | | | | | | | | | | | |
| Hematology, Chemistry | X | X | | X | | X | | | | X | | | | X | X | X | X |
| Coagulation (Prothrombin activation %, PT, aPTT and INR) | X | X | | X | | X | | | | X | | | | X | X | X | X |
| Urinalysis | X | | | | | | | | | | | | | | | | |
| HCV RNA | X | X | | X | | X | | | | X | | | | X | X | X | X |
| Viral RNA Sequencing / Phenotyping | | X | | X | | X | | | | X | | | | X | X | X | X |
| HBV DNA sample <sup>1</sup> | | | | X | | X | | | | X | | | | X | X | X | X |
| Single PK | | | | X | | X | | | | X | | | | X | | | |
| Serum or Urine Pregnancy Test <sup>m</sup> | X | X | | | | X | | | | X | | | | X | X | X | X |
| HCV Genotyping | X | | | | | | | | | | | | | | | | |
| IL28B Genotype | | X | | | | | | | | | | | | | | | |
| HCV Ab, HIV Ab, HBsAg, HBsAb, HBcAb | X | | | | | | | | | | | | | | | | |
| FibroTest <sup>®</sup> | X | | | | | | | | | | | | | | | | |
| Archive Plasma sample <sup>n</sup> | | X | | | | | | | | | | | | X | | | |
| Single Genomic sample <sup>o</sup> | | X | | | | | | | | | | | | | | | |

a Day 1 assessments must be performed prior to dosing.

b ET = early termination.

c Prior to randomization on Day 1, CPT score should be calculated using laboratory values from the local lab to verify that it is between 7-12; however, randomization will be based on CPT score at Screening.

d Vital signs include resting blood pressure, pulse, respiratory rate and temperature.

e Subjects will be required to rest in a supine position for ≥ 5 minutes prior to making a recording. The investigator (or qualified designee) should review the ECG traces recorded in real time for clinically significant abnormalities.

f Adverse events and Concomitant Medications will be collected up to 30 days after the last dose of all study drugs. In addition, records of Concomitant Medications for ascites and hepatic encephalopathy taken through posttreatment Week 24 will be collected in the eCRF.

g Health Related Quality of Life (HRQoL) Surveys (eg, SF-36, CLDQ-HCV, FACIT-F and WPAI) will be conducted for all subjects where the surveys are available at Day 1.

- h Liver imaging (eg, ultrasound or CT scan, at the discretion of the investigator) should be performed to exclude the presence of hepatocellular carcinoma (HCC) in all subjects within 4 months of Day 1.
- i Study drugs will be reconciled at every post- Day 1 visit by the investigator in order to monitor the subject's adherence with the study drugs. Subjects must be instructed to bring back all bottles of study drugs in the original container at every post- Day 1 visit through the end of treatment.
- The IWRS will provide direction on the specifics of each subject's study drug dispensing.
- k Subjects with CPT C cirrhosis at Screening should be monitored closely during treatment with SOF/VEL ± RBV. The extent and duration of monitoring is at the discretion of the Investigator, based on assessment of each individual subject, but may include daily contact with subject (or subject's family) or in-patient hospitalization. Proximity of subject's residence to the investigator's institution should be taken into consideration. The objective of this close monitoring is to facilitate prompt communication and response to adverse events that may occur.
- 1 Reflex testing done only when ALT > 2x Day 1 value in subjects who are HBsAb or HBcAb positive at Screening.
- Mall females of childbearing potential will have a serum pregnancy test at Screening. Urine pregnancy testing will occur at Day 1 and every 4 weeks through posttreatment Week 4. In addition, females of childbearing potential in the treatment group receiving RBV will have additional urine pregnancy testing every 4 weeks for a minimum of 6 months following last dose of RBV. If required by local regulations, additional pregnancy tests beyond 6 months may be added. In the event of a positive urine pregnancy result, subjects will be instructed to return to the clinic as soon as possible for a serum pregnancy test. The subject will be contacted by telephone monthly to confirm that urine pregnancy testing has been performed posttreatment and to record the outcome. Alternatively, if required by local regulations or preferred by the investigator or subject, the subject may return to the clinic for urine pregnancy tests.
- n Only for subjects who have provided separate consent for this sample and testing
- o Only for subjects who have provided separate consent for this sample and testing. This sample can be obtained at a subsequent visit if not obtained at Day 1.

Appendix 3. GSI Grading Scale for Severity of Adverse Events and Laboratory Abnormalities

Antiviral Toxicity Grading Scale Version: 01 April 2015

| | | HEMATOLOGY | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hemoglobin<br>HIV POSITIVE<br>Adult and Pediatric ≥ 57 Days | 8.5 to 10.0 g/dL<br>85 to 100 g/L | 7.5 to < 8.5 g/dL<br>75 to < 85 g/L | 6.5 to < 7.5 g/dL<br>65 to < 75 g/L | < 6.5 g/dL<br>< 65 g/L |
| HIV NEGATIVE Adult and Pediatric ≥ 57 Days | 10.0 to 10.9 g/dL<br>100 to 109 g/L<br>OR<br>Any decrease from Baseline<br>2.5 to < 3.5 g/dL<br>25 to < 35 g/L | 9.0 to < 10.0 g/dL<br>90 to < 100 g/L<br>OR<br>Any decrease from Baseline<br>3.5 to < 4.5 g/dL<br>35 to < 45 g/L | 7.0 to $<$ 9.0 g/dL<br>70 to $<$ 90 g/L<br>OR<br>Any decrease from Baseline<br>$\ge$ 4.5 g/dL<br>$\ge$ 45 g/L | < 7.0 g/dL<br>< 70 g/L |
| Infant, 36–56 Days<br>(HIV <u>POSITIVE</u> OR<br><u>NEGATIVE</u> ) | 8.5 to 9.4 g/dL<br>85 to 94 g/L | 7.0 to < 8.5 g/dL<br>70 to < 85 g/L | 6.0 to < 7.0 g/dL<br>60 to < 70 g/L | < 6.0 g/dL<br>< 60 g/L |
| Infant, 22–35 Days<br>(HIV <u>POSITIVE</u> OR<br><u>NEGATIVE</u> ) | 9.5 to 10.5 g/dL<br>95 to 105 g/L | 8.0 to < 9.5 g/dL<br>80 to < 95 g/L | 7.0 to < 8.0 g/dL<br>70 to < 80 g/L | < 7.0 g/dL<br>< 70 g/L |
| Infant, 1–21 Days<br>(HIV <u>POSITIVE</u> OR<br><u>NEGATIVE</u> ) | 12.0 to 13.0 g/dL<br>120 to 130 g/L | 10.0 to < 12.0 g/dL<br>100 to < 120 g/L | 9.0 to < 10.0 g/dL<br>90 to < 100 g/L | < 9.0 g/dL<br>< 90 g/L |
| Absolute Neutrophil Count (ANC) Adult and Pediatric, ≥ 7 Months# | 1000 to 1300/mm <sup>3</sup> 1.00 to 1.30 GI/L | 750 to < 1000/mm <sup>3</sup><br>0.75 to < 1.00 GI/L | 500 to < 750/mm <sup>3</sup><br>0.50 to < 0.75 GI/L | < 500/mm <sup>3</sup><br>< 0.50 GI/L |
| Absolute CD4+ Count HIV NEGATIVE ONLY Adult and Pediatric > 13 Years | 300 to 400/mm <sup>3</sup><br>300 to 400/μL | 200 to < 300/mm <sup>3</sup><br>200 to < 300/μL | $100 \text{ to} < 200/\text{mm}^3 \\ 100 \text{ to} < 200/\mu L$ | < 100/mm <sup>3</sup><br>< 100/μL |

| | | HEMATOLOGY | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Absolute Lymphocyte Count HIV NEGATIVE ONLY Adult and Pediatric > 13 Years | 600 to 650/mm <sup>3</sup><br>0.60 to 0.65 GI/L | 500 to < 600/mm <sup>3</sup><br>0.50 to < 0.60 GI/L | 350 to < 500/mm <sup>3</sup><br>0.35 to < 0.50 GI/L | < 350/mm <sup>3</sup><br>< 0.35 GI/L |
| Platelets | 100,000 to < 125,000/mm <sup>3</sup><br>100 to < 125 GI/L | 50,000 to < 100,000/mm <sup>3</sup><br>50 to < 100 GI/L | 25,000 to < 50,000/mm <sup>3</sup><br>25 to < 50 GI/L | < 25,000/mm <sup>3</sup><br>< 25 GI/L |
| WBCs | 2000/mm <sup>3</sup> to 2500/mm <sup>3</sup> | 1,500 to < 2,000/mm <sup>3</sup> | 1000 to < 1,500/mm <sup>3</sup> | < 1000/mm <sup>3</sup> |
| | 2.00 GI/L to 2.50 GI/L | 1.50 to < 2.00 GI/L | 1.00 to < 1.50 GI/L | < 1.00 GI/L |
| Hypofibrinogenemia | 100 to 200 mg/dL | 75 to < 100 mg/dL | 50 to < 75 mg/dL | < 50 mg/dL |
| | 1.00 to 2.00 g/L | 0.75 to < 1.00 g/L | 0.50 to < 0.75 g/L | < 0.50 g/L |
| Hyperfibrinogenemia | > ULN to 600 mg/dL | > 600 mg/dL | _ | _ |
| | > ULN to 6.0 g/L | > 6.0 g/L | _ | _ |
| Fibrin Split Product | 20 to 40 μg/mL | > 40 to 50 μg/mL | > 50 to 60 μg/mL | > 60 μg/mL |
| | 20 to 40 mg/L | > 40 to 50 mg/L | > 50 to 60 mg/L | > 60 mg/L |
| Prothrombin Time (PT) | > 1.00 to 1.25 × ULN | > 1.25 to 1.50 × ULN | > 1.50 to 3.00 × ULN | > 3.00 × ULN |
| International Normalized Ratio of prothrombin time (INR) | 1.1 to 1.5 x ULN | >1.5 to 2.0 x ULN | >2.0 to 3.0 x ULN | >3.0 x ULN |
| Activated Partial<br>Thromboplastin Time (APTT) | > 1.00 to 1.66 × ULN | > 1.66 to 2.33 × ULN | > 2.33 to 3.00 × ULN | > 3.00 × ULN |
| Methemoglobin | 5.0 to 10.0% | > 10.0 to 15.0% | > 15.0 to 20.0% | > 20.0% |

<sup>#</sup> An overlap between the Grade 1 scale and the Lab's normal range for absolute neutrophils may result for pediatric subjects. Please follow the Gilead convention of grading any result within the LLN and ULN a 0.

| | | CHEMISTRY | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hyponatremia | 130 to <lln l<="" meq="" td=""><td>125 to &lt; 130 mEq/L</td><td>121 to &lt; 125 mEq/L</td><td>&lt; 121 mEq/L</td></lln> | 125 to < 130 mEq/L | 121 to < 125 mEq/L | < 121 mEq/L |
| | 130 to <lln l<="" mmol="" td=""><td>125 to &lt; 130 mmol/L</td><td>121 to &lt; 125 mmol/L</td><td>&lt; 121 mmol/L</td></lln> | 125 to < 130 mmol/L | 121 to < 125 mmol/L | < 121 mmol/L |
| Hypernatremia | >ULN to 150 mEq/L | > 150 to 154 mEq/L | > 154 to 159 mEq/L | > 159 mEq/L |
| | >ULN to 150 mmol/L | > 150 to 154 mmol/L | > 154 to 159 mmol/L | > 159 mmol/L |
| Hypokalemia | 3.0 to <lln l<="" meq="" td=""><td>2.5 to &lt; 3.0 mEq/L</td><td>2.0 to &lt; 2.5 mEq/L</td><td>&lt; 2.0 mEq/L</td></lln> | 2.5 to < 3.0 mEq/L | 2.0 to < 2.5 mEq/L | < 2.0 mEq/L |
| Adult and Pediatric<br>≥1 Year | 3.0 to <lln l<="" mmol="" td=""><td>2.5 to &lt; 3.0 mmol/L</td><td>2.0 to &lt; 2.5 mmol/L</td><td>&lt; 2.0 mmol/L</td></lln> | 2.5 to < 3.0 mmol/L | 2.0 to < 2.5 mmol/L | < 2.0 mmol/L |
| Infant <1 Year | 3.0 to 3.4 mEq/L<br>3.0 to 3.4 mmol/L | 2.5 to < 3.0 mEq/L<br>2.5 to <3.0 mmolL | 2.0 to < 2.5 mEq/L<br>2.0 to <2.5 mmolL | < 2.0 mEq/L<br><2.0 mmolL |
| Hyperkalemia<br>Adult and Pediatric<br>≥ 1 Year | 5.6 to 6.0 mEq/L<br>5.6 to 6.0 mmol/L | > 6.0 to 6.5 mEq/L<br>> 6.0 to 6.5 mmol/L | > 6.5 to 7.0 mEq/L<br>> 6.5 to 7.0 mmol/L | > 7.0 mEq/L<br>> 7.0 mmol/L |
| Infant <1 Year | >ULN to 6.0 mEq/L<br>>ULN to 6.0 mmol/L | > 6.0 to 6.5 mEq/L<br>> 6.0 to 6.5 mmol/L | > 6.5 to 7.0 mEq/L<br>> 6.5 to 7.0 mmol/L | > 7.0 mEq/L<br>> 7.0 mmol/L |
| Hypoglycemia Adult and Pediatric ≥ 1 Month | 55 to 64 mg/dL<br>3.03 to 3.58 mmol/L | 40 to < 55 mg/dL<br>2.20 to < 3.03 mmol/L | 30 to < 40 mg/dL<br>1.64 to < 2.20 mmol/L | < 30 mg/dL<br>< 1.64 mmol/L |
| Infant, < 1 Month | 50 to 54 mg/dL<br>2.8 to 3.0 mmol/L | 40 to < 50 mg/dL<br>2.2 to < 2.8 mmol/L | 30 to < 40 mg/dL<br>1.7 to < 2.2 mmol/L | < 30 mg/dL<br>< 1.7 mmol/L |
| Hyperglycemia, Nonfasting | 116 to 160 mg/dL | > 160 to 250 mg/dL | > 250 to 500 mg/dL | > 500 mg/dL |
| | 6.42 to 8.91 mmol/L | > 8.91 to 13.90 mmol/L | > 13.90 to 27.79 mmol/L | > 27.79 mmol/L |
| Hyperglycemia, Fasting | 110 to 125 mg/dL<br>6.08 to 6.96 mmol/L | >125 to 250 mg/dL<br>>6.96 to 13.90 mmol/L | >250 to 500 mg/dL<br>>13.90 to 27.79 mmol/L | >500 mg/dL<br>>27.79 mmol/L |

| | | CHEMISTRY | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypocalcemia (corrected for albumin if appropriate*) Adult and Pediatric ≥2 Years | 7.8 <lln dl<br="" mg="">1.94 to <lln l<="" mmol="" td=""><td>7.0 to &lt; 7.8 mg/dL<br/>1.74 to &lt; 1.94 mmol/L</td><td>6.1 to &lt; 7.0 mg/dL<br/>1.51 to &lt; 1.74 mmol/L</td><td>&lt; 6.1 mg/dL<br/>&lt; 1.51 mmol/L</td></lln></lln> | 7.0 to < 7.8 mg/dL<br>1.74 to < 1.94 mmol/L | 6.1 to < 7.0 mg/dL<br>1.51 to < 1.74 mmol/L | < 6.1 mg/dL<br>< 1.51 mmol/L |
| Pediatric ≥7 days -2 Years | 7.8 to 8.4 mg/dL<br>1.94 to 2.10 mmol/L | 7.0 to <7.8 mg/dL<br>1.74 to <1.94 mmolL | 6.1 to <7.0 mg/dL<br>1.51 to < 1.74 mmolL | < 6.1 mg/dL<br>< 1.51 mmol/L |
| Infant, < 7 Days | 6.5 to 7.5 mg/dL<br>1.61 to 1.88 mmol/L | 6.0 to < 6.5 mg/dL<br>1.49 to < 1.61 mmol/L | 5.5 to < 6.0 mg/dL<br>1.36 to < 1.49 mmol/L | < 5.5 mg/dL<br>< 1.36 mmol/L |
| Hypercalcemia (corrected for albumin if appropriate*) Adult and Pediatric ≥ 7 Days | >ULN to 11.5 mg/dL<br>>ULN to 2.88 mmol/L | > 11.5 to 12.5 mg/dL<br>> 2.88 to 3.13 mmol/L | > 12.5 to 13.5 mg/dL<br>> 3.13 to 3.38 mmol/L | > 13.5 mg/dL<br>> 3.38 mmol/L |
| Infant, < 7 Days | 11.5 to 12.4 mg/dL<br>2.86 to 3.10 mmol/L | > 12.4 to 12.9 mg/dL<br>> 3.10 to 3.23 mmol/L | > 12.9 to 13.5 mg/dL<br>> 3.23 to 3.38 mmol/L | > 13.5 mg/dL<br>> 3.38 mmol/L |
| Hypocalcemia (ionized) | 3.0 mg/dL to < LLN | 2.5 to < 3.0 mg/dL | 2.0 to < 2.5 mg/dL | < 2.0 mg/dL |
| | 0.74 mmol/L to < LLN | 0.62 to < 0.74 mmol/L | 0.49 to < 0.62 mmol/L | < 0.49 mmol/L |
| Hypercalcemia (ionized) | > ULN to 6.0 mg/dL | > 6.0 to 6.5 mg/dL | > 6.5 to 7.0 mg/dL | > 7.0 mg/dL |
| | > ULN to 1.50 mmol/L | > 1.50 to 1.63 mmol/L | > 1.63 to 1.75 mmol/L | > 1.75 mmol/L |
| Hypomagnesemia | 1.40 to <lln dl<br="" mg="">1.2 to <lln l<="" meq="" td=""><td>1.04 to &lt; 1.40 mg/dL<br/>0.9 to &lt; 1.2 mEq/L</td><td>0.67 to &lt; 1.04 mg/dL<br/>0.6 to &lt; 0.9 mEq/L</td><td>&lt; 0.67 mg/dL<br/>&lt; 0.6 mEq/L</td></lln></lln> | 1.04 to < 1.40 mg/dL<br>0.9 to < 1.2 mEq/L | 0.67 to < 1.04 mg/dL<br>0.6 to < 0.9 mEq/L | < 0.67 mg/dL<br>< 0.6 mEq/L |
| | 0.58 to <lln l<="" mmol="" td=""><td>0.43 to &lt; 0.58 mmol/L</td><td>0.28 to &lt; 0.43 mmol/L</td><td>&lt; 0.28 mmol/L</td></lln> | 0.43 to < 0.58 mmol/L | 0.28 to < 0.43 mmol/L | < 0.28 mmol/L |

| | | CHEMISTRY | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hypophosphatemia Adult and Pediatric > 14 Years | 2.0 to < LLN mg/dL<br>0.63 to < LLN mmol/L | 1.5 to < 2.0 mg/dL<br>0.47 to < 0.63 mmol/L | 1.0 to < 1.5 mg/dL<br>0.31 to < 0.47 mmol/L | < 1.0 mg/dL<br>< 0.31 mmol/L |
| Pediatric 1 Year–14 Years | 3.0 to <lln dl<br="" mg="">0.96 to <lln l<="" mmol="" td=""><td>2.5 to &lt; 3.0 mg/dL<br/>0.80 to &lt; 0.96 mmol/L</td><td>1.5 to &lt; 2.5 mg/dL<br/>0.47 to &lt; 0.80 mmol/L</td><td>&lt; 1.5 mg/dL<br/>&lt; 0.47 mmol/L</td></lln></lln> | 2.5 to < 3.0 mg/dL<br>0.80 to < 0.96 mmol/L | 1.5 to < 2.5 mg/dL<br>0.47 to < 0.80 mmol/L | < 1.5 mg/dL<br>< 0.47 mmol/L |
| Pediatric < 1 Year | 3.5 to <lln dl<br="" mg="">1.12 to <lln l<="" mmol="" td=""><td>2.5 to &lt; 3.5 mg/dL<br/>0.80 to &lt; 1.12 mmol/L</td><td>1.5 to &lt; 2.5 mg/dL<br/>0.47 to &lt; 0.80 mmol/L</td><td>&lt; 1.5 mg/dL<br/>&lt; 0.47 mmol/L</td></lln></lln> | 2.5 to < 3.5 mg/dL<br>0.80 to < 1.12 mmol/L | 1.5 to < 2.5 mg/dL<br>0.47 to < 0.80 mmol/L | < 1.5 mg/dL<br>< 0.47 mmol/L |
| Hyperbilirubinemia Adult and Pediatric > 14 Days | > 1.0 to 1.5 × ULN | > 1.5 to 2.5 × ULN | > 2.5 to 5.0 × ULN | > 5.0 × ULN |
| Infant, ≤ 14 Days (non-hemolytic) | NA | 20.0 to 25.0 mg/dL<br>342 to 428 μmol/L | > 25.0 to 30.0 mg/dL<br>> 428 to 513 μmol/L | > 30.0 mg/dL<br>> 513 µmol/L |
| Infant, ≤ 14 Days (hemolytic) | NA | NA | 20.0 to 25.0 mg/dL<br>342 to 428 μmol/L | > 25.0 mg/dL<br>> 428 µmol/L |
| Blood Urea Nitrogen | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Hyperuricemia | >ULN to 10.0 mg/dL | > 10.0 to 12.0 mg/dL | > 12.0 to 15.0 mg/dL | > 15.0 mg/dL |
| | >ULN to 597 μmol/L | > 597 to 716 μmol/L | > 716 to 895 μmol/L | > 895 μmol/L |
| Hypouricemia Adult and Pediatric | 1.5 mg/dL to < LLN<br>87 μmol/L to < LLN | 1.0 to < 1.5 mg/dL<br>57 to < 87 μmol/L | 0.5 to < 1.0 mg/dL<br>27 to < 57 μmol/L | < 0.5 mg/dL<br>< 27 μmol/L |
| ≥1 year<br>Infant <1 Year | N/A | 1.0 mg/dl to <lln<br>57 μmol to <lln< td=""><td>0.5 to &lt; 1.0 mg/dL<br/>27 to &lt; 57 μmol/L</td><td>&lt; 0.5 mg/dL<br/>&lt; 27 μmol/L</td></lln<></lln<br> | 0.5 to < 1.0 mg/dL<br>27 to < 57 μmol/L | < 0.5 mg/dL<br>< 27 μmol/L |
| Creatinine** | > 1.50 to 2.00 mg/dL<br>> 133 to 177 μmol/L | > 2.00 to 3.00 mg/dL<br>> 177 to 265 μmol/L | > 3.00 to 6.00 mg/dL<br>> 265 to 530 μmol/L | > 6.00 mg/dL<br>> 530 μmol/L |

| | | CHEMISTRY | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Bicarbonate | 16.0 mEq/L to < LLN | 11.0 to < 16.0 mEq/L | 8.0 to < 11.0 mEq/L | < 8.0 mEq/L |
| Adult and Pediatric<br>≥ 4 Years | 16.0 mmol/L to < LLN | 11.0 to < 16.0 mmol/L | 8.0 to < 11.0 mmol/L | < 8.0 mmol/L |
| Pediatric < 4 Years | NA | 11.0 mEq/Lto <lln< td=""><td>8.0 to &lt; 11.0 mEq/L</td><td>&lt; 8.0 mEq/L</td></lln<> | 8.0 to < 11.0 mEq/L | < 8.0 mEq/L |
| | | 11.0 mmol/L to <lln< td=""><td>8.0 to &lt; 11.0 mmol/L</td><td>&lt; 8.0 mmol/L</td></lln<> | 8.0 to < 11.0 mmol/L | < 8.0 mmol/L |
| Triglycerides<br>(Fasting) | NA | 500 to 750 mg/dL<br>5.64–8.47 mmol/L | > 750 to 1200 mg/dL<br>> 8.47–13.55 mmol/L | > 1200 mg/dL<br>> 13.55 mmol/L |
| LDL (Fasting) | 130 to 160 mg/dL | >160 to 190 mg/dL | > 190 mg/dL | NA |
| Adult | 3.35 to 4.15 mmol/L | >4.15 to 4.92 mmol/L | >4.92 mmol/L | |
| LDL (Fasting) | 110 to 130 mg/dL | >130 to 190 mg/dL | > 190 mg/dL | NA |
| Pediatric >2 to <18 years | 2.84 to 3.37 mmol/L | >3.37 to 4.92 mmol/L | >4.92 mmol/L | |
| Hypercholesterolemia | 200 to 239 mg/dL | > 239 to 300 mg/dL | > 300 mg/dL | NA |
| (Fasting) | 5.16 to 6.19 mmol/L | > 6.19 to 7.77 mmol/L | > 7.77 mmol/L | |
| Pediatric < 18 Years | 170 to 199 mg/dL<br>4.39 to 5.15 mmol/L | > 199 to 300 mg/dL<br>> 5.15 to 7.77 mmol/L | > 300 mg/dL<br>> 7.77 mmol/L | NA |
| Creatine Kinase | $3.0 \text{ to} < 6.0 \times \text{ULN}$ | 6.0 to < 10.0 × ULN | 10.0 to < 20.0 × ULN | ≥ 20.0 × ULN |

Calcium should be corrected for albumin if albumin is < 4.0 g/dL

An overlap between the Grade 1 scale and the Lab's normal range for creatinine may result for Male subjects >70 yrs. Please follow the Gilead convention of grading any result within the LLN and ULN a 0.

| | | ENZYMES | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| AST (SGOT) | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| ALT (SGPT) | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| GGT | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Alkaline Phosphatase | 1.25 to 2.50 × ULN | > 2.50 to 5.00 × ULN | > 5.00 to 10.00 × ULN | > 10.00 × ULN |
| Total Amylase | > 1.0 to 1.5 × ULN | > 1.5 to 2.0 × ULN | > 2.0 to 5.0 × ULN | > 5.0 × ULN |
| Pancreatic Amylase | > 1.0 to 1.5 × ULN | > 1.5 to 2.0 × ULN | > 2.0 to 5.0 × ULN | > 5.0 × ULN |
| Lipase | > 1.0 to 1.5 × ULN | > 1.5 to 3.0 × ULN | > 3.0 to 5.0 × ULN | > 5.0 × ULN |
| Albumin Pediatrics <16 years | - | 2.0 to < LLN g/dL<br>20 to < LLN g/L | < 2.0 g/dL<br>< 20 g/L | NA |
| ≥ 16 years | 3.0 g/dL to < LLN<br>30 g/L to < LLN | 2.0 to < 3.0 g/dL<br>20 to < 30 g/L | < 2.0 g/dL<br>< 20 g/L | NA |

| | | URINALYSIS | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Hematuria (Dipstick) | 1+ | 2+ | 3-4+ | NA |
| Hematuria (Quantitative) See Note below Females | >ULN - 10 RBC/HPF | > 10-75 RBC/HPF | > 75 RBC/HPF | NA |
| Males | 6-10 RBC/HPF | > 10-75 RBC/HPF | > 75 RBC/HPF | NA |
| Proteinuria (Dipstick) | 1+ | 2–3+ | 4+ | NA |
| Proteinuria, 24 Hour Collection Adult and Pediatric ≥ 10 Years | 200 to 999 mg/24 h | >999 to 1999 mg/24 h | >1999 to 3500 mg/24 h | > 3500 mg/24 h |
| Pediatric > 3 Mo to<br>< 10 Years | 201 to 499 mg/m <sup>2</sup> /24 h | >499 to 799 mg/m <sup>2</sup> /24 h | >799 to 1000 mg/m <sup>2</sup> /24 h | > 1000 mg/ m <sup>2</sup> /24 h |
| Glycosuria (Dipstick) | 1+ | 2-3+ | 4+ | NA |

#### Notes:

- Toxicity grades for Quantitative and Dipstick Hematuria will be assigned by Covance Laboratory, however for other laboratories, toxicity grades will only be assigned to Dipstick Hematuria.
- With the exception of lipid tests, any graded laboratory test with a result that is between the LLN and ULN should be assigned Grade 0.
- If the severity of a clinical AE could fall under either one of two grades (e.g., the severity of an AE could be either Grade 2 or Grade 3), select the higher of the two grades for the AE.

| | CARDIOVASCULAR | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Cardiac Arrhythmia (general)<br>(By ECG or physical exam) | Asymptomatic AND No intervention indicated | Asymptomatic AND Non-<br>urgent medical intervention<br>indicated | Symptomatic, non-life-<br>threatening AND Non-<br>urgent medical intervention<br>indicated | Life-threatening arrhythmia<br>OR Urgent intervention<br>indicated |
| Cardiac-ischemia/Infarction | NA | NA | Symptomatic ischemia (stable angina) OR Testing consistent with ischemia | Unstable angina OR Acute myocardial infarction |
| Hemorrhage (significant acute blood loss) | NA | Symptomatic AND No transfusion indicated | Symptomatic AND Transfusion of ≤ 2 units packed RBCs (for children ≤ 10 cc/kg) indicated | Life-threatening hypotension<br>OR Transfusion of > 2 units<br>packed RBCs indicated (for<br>children ≤ 10 cc/kg) indicated |
| Hypertension (with repeat testing at same visit) | 140–159 mmHg systolic<br>OR<br>90–99 mmHg diastolic | > 159–179 mmHg systolic<br>OR<br>> 99–109 mmHg diastolic | > 179 mmHg systolic<br>OR<br>> 109 mmHg diastolic | Life-threatening consequences<br>(eg, malignant hypertension)<br>OR Hospitalization (other than<br>ER visit) indicated |
| Pediatric ≤ 17 Years (with repeat testing at same visit) | NA | 91st–94th percentile adjusted<br>for age, height, and gender<br>(systolic and/or diastolic) | ≥ 95th percentile adjusted for age, height, and gender (systolic and/or diastolic) | Life-threatening consequences (eg, malignant hypertension) OR Hospitalization indicated (other than emergency room visit) |
| Hypotension | NA | Symptomatic, corrected with oral fluid replacement | Symptomatic, IV fluids indicated | Shock requiring use of vasopressors or mechanical assistance to maintain blood pressure |
| Pericardial Effusion | Asymptomatic, small effusion requiring no intervention | Asymptomatic, moderate or larger effusion requiring no intervention | Effusion with non-life-<br>threatening physiologic<br>consequences OR Effusion<br>with nonurgent intervention<br>indicated | Life-threatening consequences<br>(eg, tamponade) OR Urgent<br>intervention indicated |

| | CARDIOVASCULAR | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Prolonged PR Interval | PR interval 0.21 to 0.25 sec | PR interval > 0.25 sec | Type II 2nd degree AV<br>block OR Ventricular pause<br>> 3.0 sec | Complete AV block |
| Pediatric ≤ 16 Years | 1st degree AV block<br>(PR > normal for age and rate) | Type I 2nd degree AV block | Type II 2nd degree AV block | Complete AV block |
| Prolonged QTc | Asymptomatic, QTc interval 0.45 to 0.47 sec OR Increase interval < 0.03 sec above baseline | Asymptomatic, QTc interval 0.48 to 0.49 sec OR Increase in interval 0.03 to 0.05 sec above baseline | Asymptomatic, QTc interval ≥ 0.50 sec OR Increase in interval ≥ 0.06 sec above baseline | Life-threatening<br>consequences, eg, Torsade de<br>pointes or other associated<br>serious ventricular<br>dysrhythmia |
| Pediatric ≤ 16 Years | Asymptomatic, QTc interval 0.450 to 0.464 sec | Asymptomatic, QTc interval 0.465 to 0.479 sec | Asymptomatic, QTc interval ≥ 0.480 sec | Life-threatening<br>consequences, eg, Torsade de<br>pointes or other associated<br>serious ventricular<br>dysrhythmia |
| Thrombosis/Embolism | NA | Deep vein thrombosis AND<br>No intervention indicated (eg,<br>anticoagulation, lysis filter,<br>invasive procedure) | Deep vein thrombosis AND<br>Intervention indicated (eg,<br>anticoagulation, lysis filter,<br>invasive procedure) | Embolic event (eg, pulmonary embolism, life-threatening thrombus) |
| Vasovagal Episode (associated with a procedure of any kind) | Present without loss of consciousness | Present with transient loss of consciousness | NA | NA |
| Ventricular Dysfunction<br>(congestive heart failure,<br>CHF) | NA | Asymptomatic diagnostic finding AND intervention indicated | New onset with symptoms<br>OR Worsening symptomatic<br>CHF | Life-threatening CHF |

| RESPIRATORY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Bronchospasm (acute) | FEV1 or peak flow reduced to 70% to 80% | FEV1 or peak flow 50% to 69% | FEV1 or peak flow 25% to 49% | Cyanosis OR FEV1 or peak flow < 25% OR Intubation |
| Dyspnea or Respiratory<br>Distress | Dyspnea on exertion with no or minimal interference with usual social & functional activities | Dyspnea on exertion causing greater than minimal interference with usual social & functional activities | Dyspnea at rest causing inability to perform usual social & functional activities | Respiratory failure with ventilatory support indicated |
| Pediatric < 14 Years | Wheezing OR minimal increase in respiratory rate for age | Nasal flaring OR Intercostal retractions OR Pulse oximetry 90% to 95% | Dyspnea at rest causing inability to perform usual social & functional activities OR Pulse oximetry < 90% | Respiratory failure with ventilatory support indicated |

| OCULAR/VISUAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Uveitis | Asymptomatic but detectable on exam | Symptomatic anterior uveitis OR<br>Medical intervention indicated | Posterior or pan-uveitis OR<br>Operative intervention<br>indicated | Disabling visual loss in affected eye(s) |
| Visual Changes (from baseline) | Visual changes causing no or minimal interference with usual social & functional activities | Visual changes causing greater than minimal interference with usual social & functional activities | Visual changes causing inability to perform usual social & functional activities | Disabling visual loss in affected eye(s) |

| SKIN | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alopecia | Thinning detectable by study participant or caregiver (for disabled adults) | Thinning or patchy hair loss detectable by health care provider | Complete hair loss | NA |
| Cutaneous Reaction – Rash | Localized macular rash | Diffuse macular,<br>maculopapular, or<br>morbilliform rash OR Target<br>lesions | Diffuse macular,<br>maculopapular, or morbilliform<br>rash with vesicles or limited<br>number of bullae OR<br>Superficial ulcerations of<br>mucous membrane limited to<br>one site | Extensive or generalized<br>bullous lesions OR<br>Stevens-Johnson syndrome<br>OR Ulceration of mucous<br>membrane involving two<br>or more distinct mucosal<br>sites OR Toxic epidermal<br>necrolysis (TEN) |
| Hyperpigmentation | Slight or localized | Marked or generalized | NA | NA |
| Hypopigmentation | Slight or localized | Marked or generalized | NA | NA |
| Pruritis (itching – no skin lesions) (See also Injection Site Reactions: Pruritis associated with injection) | Itching causing no or minimal interference with usual social & functional activities | Itching causing greater than minimal interference with usual social & functional activities | Itching causing inability to perform usual social & functional activities | NA |

| | GASTROINTESTINAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Anorexia | Loss of appetite without decreased oral intake | Loss of appetite associated with decreased oral intake without significant weight loss | Loss of appetite associated with significant weight loss | Life-threatening consequences<br>OR Aggressive intervention<br>indicated [eg, tube feeding or<br>total parenteral nutrition] |
| Ascites | Asymptomatic | Symptomatic AND Intervention indicated (eg, diuretics or therapeutic paracentesis) | Symptomatic despite intervention | Life-threatening consequences |
| Cholecystitis | NA | Symptomatic AND Medical intervention indicated | Radiologic, endoscopic, or operative intervention indicated | Life-threatening consequences (eg, sepsis or perforation) |
| Constipation | NA | Persistent constipation requiring regular use of dietary modifications, laxatives, or enemas | Obstipation with manual evacuation indicated | Life-threatening consequences (eg, obstruction) |
| Diarrhea Adult and Pediatric ≥1 Year | Transient or intermittent episodes of unformed stools OR Increase of ≤ 3 stools over baseline/24 hr | Persistent episodes of unformed to watery stools OR Increase of 4–6 stools over baseline per 24 hrs. | Bloody diarrhea OR Increase<br>of ≥ 7 stools per 24-hour<br>period OR IV fluid<br>replacement indicated | Life-threatening consequences (eg, hypotensive shock) |
| Pediatric < 1 Year | Liquid stools (more unformed than usual) but usual number of stools | Liquid stools with increased<br>number of stools OR Mild<br>dehydration | Liquid stools with moderate dehydration | Liquid stools resulting in<br>severe dehydration with<br>aggressive rehydration<br>indicated OR Hypotensive<br>shock |
| Dysphagia-Odynophagia | Symptomatic but able to eat usual diet | Symptoms causing altered dietary intake without medical intervention indicated | Symptoms causing severely altered dietary intake with medical intervention indicated | Life-threatening reduction in oral intake |

| | GASTROINTESTINAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Mucositis/Stomatitis<br>(clinical exam)<br>See also Proctitis,<br>Dysphagia-Odynophagia | Erythema of the mucosa | Patchy pseudomembranes or ulcerations | Confluent pseudomembranes or ulcerations OR Mucosal bleeding with minor trauma | Tissue necrosis OR Diffuse<br>spontaneous mucosal bleeding<br>OR Life-threatening<br>consequences (eg, aspiration,<br>choking) |
| Nausea | Transient (< 24 hours) or intermittent nausea with no or minimal interference with oral intake | Persistent nausea resulting in decreased oral intake for 24-48 hours | Persistent nausea resulting in minimal oral intake for > 48 hours OR Aggressive rehydration indicated (eg, IV fluids) | Life-threatening consequences (eg, hypotensive shock) |
| Pancreatitis | NA | Symptomatic AND<br>Hospitalization not indicated<br>(other than ER visit) | Symptomatic AND<br>Hospitalization indicated<br>(other than ER visit) | Life-threatening consequences<br>(eg, sepsis, circulatory failure,<br>hemorrhage) |
| Proctitis (functional-<br>symptomatic)<br>Also see Mucositis/<br>Stomatitis for Clinical<br>Exam | Rectal discomfort AND No intervention indicated | Symptoms causing greater than minimal interference with usual social & functional activities OR Medical intervention indicated | Symptoms causing inability to perform usual social/ functional activities OR Operative intervention indicated | Life-threatening consequences (eg, perforation) |
| Vomiting | Transient or intermittent vomiting with no or minimal interference with oral intake | Frequent episodes of vomiting with no or mild dehydration | Persistent vomiting resulting in orthostatic hypotension OR Aggressive rehydration indicated | Life-threatening consequences (eg, hypotensive shock) |

| NEUROLOGICAL | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Alteration in<br>Personality-Behavior or in<br>Mood (eg, agitation,<br>anxiety, depression, mania,<br>psychosis) | Alteration causing no or minimal interference with usual social & functional activities | Alteration causing greater than minimal interference with usual social & functional activities | Alteration causing inability to perform usual social & functional activities | Behavior potentially harmful<br>to self or others<br>(eg, suicidal/homicidal<br>ideation or attempt, acute<br>psychosis) OR Causing<br>inability to perform basic<br>self-care functions |
| Altered Mental Status For Dementia, see Cognitive and Behavioral/Attentional Disturbance (including dementia and ADD) | Changes causing no or minimal interference with usual social & functional activities | Mild lethargy or somnolence<br>causing greater than minimal<br>interference with usual social<br>& functional activities | Confusion, memory impairment, lethargy, or somnolence causing inability to perform usual social & functional activities | Delirium OR obtundation, OR coma |
| Ataxia | Asymptomatic ataxia detectable on exam OR Minimal ataxia causing no or minimal interference with usual social & functional activities | Symptomatic ataxia causing greater than minimal interference with usual social & functional activities | Symptomatic ataxia causing inability to perform usual social & functional activities | Disabling ataxia causing inability to perform basic self-care functions |
| Cognitive and Behavioral/Attentional Disturbance (including dementia and Attention Deficit Disorder) | Disability causing no or<br>minimal interference with<br>usual social & functional<br>activities OR Specialized<br>resources not indicated | Disability causing greater than minimal interference with usual social & functional activities OR Specialized resources on part-time basis indicated | Disability causing inability to perform usual social & functional activities OR Specialized resources on a full-time basis indicated | Disability causing inability to perform basic self-care functions OR Institutionalization indicated |
| CNS Ischemia (acute) | NA | NA | Transient ischemic attack | Cerebral vascular accident (CVA, stroke) with neurological deficit |

| | NEUROLOGICAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Developmental delay – Pediatric ≤ 16 Years | Mild developmental delay, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting | Moderate developmental<br>delay, either motor or<br>cognitive, as determined by<br>comparison with a<br>developmental screening tool<br>appropriate for the setting | Severe developmental delay, either motor or cognitive, as determined by comparison with a developmental screening tool appropriate for the setting | Developmental regression,<br>either motor or cognitive, as<br>determined by comparison<br>with a developmental<br>screening tool appropriate for<br>the setting |
| Headache | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Symptoms causing inability to perform basic self-care functions OR Hospitalization indicated (other than ER visit) OR Headache with significant impairment of alertness or other neurologic function |
| Insomnia | NA | Difficulty sleeping causing greater than minimal interference with usual social/functional activities | Difficulty sleeping causing inability to perform usual social & functional activities | Disabling insomnia causing inability to perform basic self-care functions |
| Neuromuscular Weakness<br>(including myopathy &<br>neuropathy) | Asymptomatic with decreased strength on exam OR Minimal muscle weakness causing no or minimal interference with usual social & functional activities | Muscle weakness causing greater than minimal interference with usual social & functional activities | Muscle weakness causing inability to perform usual social & functional activities | Disabling muscle weakness<br>causing inability to perform<br>basic self-care functions OR<br>Respiratory muscle weakness<br>impairing ventilation |
| Neurosensory Alteration<br>(including paresthesia and<br>painful neuropathy) | Asymptomatic with sensory alteration on exam or minimal paresthesia causing no or minimal interference with usual social & functional activities | Sensory alteration or paresthesia causing greater than minimal interference with usual social & functional activities | Sensory alteration or paresthesia causing inability to perform usual social & functional activities | Disabling sensory alteration or<br>paresthesia causing inability to<br>perform basic self-care<br>functions |

| | NEUROLOGICAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Seizure: (new onset) | NA | 1 seizure | 2–4 seizures | Seizures of any kind that are prolonged, repetitive (eg, status epilepticus), or difficult to control (eg, refractory epilepsy) |
| Seizure: (pre-existing) For Worsening of Existing Epilepsy the Grades Should Be Based on an Increase from Previous Level of Control to Any of These Levels | NA | Increased frequency of pre-<br>existing seizures (non-<br>repetitive) without change in<br>seizure character OR<br>infrequent breakthrough<br>seizures while on stable meds<br>in a previously controlled<br>seizure disorder | Change in seizure character<br>from baseline either in<br>duration or quality (eg,<br>severity or focality) | Seizures of any kind that are prolonged, repetitive (eg, status epilepticus), or difficult to control (eg, refractory epilepsy) |
| Seizure - Pediatric < 18 Years | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting<br>< 5 minutes with < 24 hours<br>post ictal state | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting<br>5-20 minutes with<br>< 24 hours post ictal state | Seizure, generalized onset<br>with or without secondary<br>generalization, lasting<br>> 20 minutes | Seizure, generalized onset<br>with or without secondary<br>generalization, requiring<br>intubation and sedation |
| Syncope (not associated with a procedure) | NA | Present | NA | NA |
| Vertigo | Vertigo causing no or<br>minimal interference with<br>usual social & functional<br>activities | Vertigo causing greater than minimal interference with usual social & functional activities | Vertigo causing inability to perform usual social & functional activities | Disabling vertigo causing inability to perform basic self-care functions |

| | MUSCULOSKELETAL | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Arthralgia<br>See also Arthritis | Joint pain causing no or minimal interference with usual social & functional activities | Joint pain causing greater than minimal interference with usual social & functional activities | Joint pain causing inability to perform usual social & functional activities | Disabling joint pain causing inability to perform basic self-care functions |
| Arthritis<br>See also Arthralgia | Stiffness or joint swelling causing no or minimal interference with usual social & functional activities | Stiffness or joint swelling causing greater than minimal interference with usual social & functional activities | Stiffness or joint swelling causing inability to perform usual social & functional activities | Disabling joint stiffness or<br>swelling causing inability to<br>perform basic self-care<br>functions |
| Bone Mineral Loss | BMD t-score or z-score<br>-2.5 to -1.0 | BMD t-score or z-score < -2.5 | Pathological fracture<br>(including loss of vertebral<br>height) | Pathologic fracture causing life-threatening consequences |
| Pediatric < 21 Years | BMD z-score<br>-2.5 to -1.0 | BMD z-score < -2.5 | Pathological fracture<br>(including loss of vertebral<br>height) | Pathologic fracture causing life-threatening consequences |
| Myalgia<br>(non-injection site) | Muscle pain causing no or minimal interference with usual social & functional activities | Muscle pain causing greater than minimal interference with usual social & functional activities | Muscle pain causing inability to perform usual social & functional activities | Disabling muscle pain causing inability to perform basic self-care functions |
| Osteonecrosis | NA | Asymptomatic with radiographic findings AND No operative intervention indicated | Symptomatic bone pain with radiographic findings OR Operative intervention indicated | Disabling bone pain with radiographic findings causing inability to perform basic self-care functions |

| SYSTEMIC | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Acute Systemic Allergic<br>Reaction | Localized urticaria<br>(wheals) with no medical<br>intervention indicated | Localized urticaria with medical intervention indicated OR Mild angioedema with no medical intervention indicated | Generalized urticaria OR<br>Angioedema with medical<br>intervention indicated OR<br>Symptomatic mild<br>bronchospasm | Acute anaphylaxis OR Life-<br>threatening bronchospasm OR<br>laryngeal edema |
| Chills | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | NA |
| Fatigue<br>Malaise | Symptoms causing no or minimal interference with usual social & functional activities | Symptoms causing greater than minimal interference with usual social & functional activities | Symptoms causing inability to perform usual social & functional activities | Incapacitating fatigue/malaise symptoms causing inability to perform basic self-care functions |
| Fever (nonaxillary) | 37.7°C to 38.6°C<br>99.8°F to 101.5°F | 38.7°C to 39.3°C<br>101.6°F to 102.8°F | 39.4°C to 40.5°C<br>102.9°F to 104.9°F | > 40.5°C<br>> 104.9°F |
| Pain- Indicate Body Site<br>See also Injection Site<br>Pain, Headache,<br>Arthralgia, and Myalgia | Pain causing no or<br>minimal interference with<br>usual social & functional<br>activities | Pain causing greater than minimal interference with usual social & functional activities | Pain causing inability to perform usual social & functional activities | Disabling pain causing inability to perform basic self-care functions OR Hospitalization (other than ER visit) indicated |
| Unintentional Weight<br>Loss | NA | 5% to 9% loss in body weight from baseline | 10% to 19% loss in body<br>weight from baseline | ≥ 20% loss in body weight<br>from baseline OR Aggressive<br>intervention indicated<br>[eg, tube feeding or total<br>parenteral nutrition] |

| INJECTION SITE REACTION | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Injection Site Pain (pain<br>without touching)<br>Or Tenderness (pain when<br>area is touched) | Pain/tenderness causing no or minimal limitation of use of limb | Pain/tenderness limiting use of limb OR Pain/tenderness causing greater than minimal interference with usual social & functional activities | Pain/tenderness causing inability to perform usual social & functional activities | Pain/tenderness causing inability<br>to perform basic self-care<br>function OR Hospitalization<br>(other than ER visit) indicated<br>for management of<br>pain/tenderness |
| Injection Site Reaction (Localized), > 15 Years | Erythema OR Induration<br>of $5 \times 5$ cm to $9 \times 9$ cm (or<br>$25-81 \times \text{cm}^2$ ) | Erythema OR Induration OR<br>Edema > 9 cm any diameter<br>(or > 81 cm <sup>2</sup> ) | Ulceration OR Secondary<br>infection OR Phlebitis OR<br>Sterile abscess OR Drainage | Necrosis (involving dermis and deeper tissue) |
| Pediatric ≤ 15 Years | Erythema OR Induration<br>OR Edema present but<br>≤ 2.5 cm diameter | Erythema OR Induration<br>OR Edema > 2.5 cm<br>diameter but < 50% surface<br>area of the extremity<br>segment (eg, upper<br>arm/thigh) | Erythema OR Induration OR Edema involving ≥ 50% surface area of the extremity segment (eg, upper arm/thigh) OR Ulceration OR Secondary infection OR Phlebitis OR Sterile abscess OR Drainage | Necrosis (involving dermis and deeper tissue) |
| Pruritis Associated with<br>Injection<br>See also Skin: Pruritis<br>(itching—no skin lesions) | Itching localized to injection site AND Relieved spontaneously or with < 48 h treatment | Itching beyond the injection site but not generalized OR Itching localized to injection site requiring ≥ 48 h treatment | Generalized itching causing inability to perform usual social & functional activities | NA |

| ENDOCRINE/METABOLIC | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Lipodystrophy (eg, back of neck, breasts, abdomen) | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious changes on casual visual inspection | NA |
| Diabetes Mellitus | NA | New onset without need to initiate medication OR Modification of current meds to regain glucose control | New onset with initiation of indicated med OR Diabetes uncontrolled despite treatment modification | Life-threatening consequences (eg, ketoacidosis, hyperosmolar non-ketotic coma) |
| Gynecomastia | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious on casual visual inspection | NA |
| Hyperthyroidism | Asymptomatic | Symptomatic causing greater than minimal interference with usual social & functional activities OR Thyroid suppression therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (eg, thyroid storm) |
| Hypothyroidism | Asymptomatic | Symptomatic causing greater than minimal interference with usual social & functional activities OR Thyroid replacement therapy indicated | Symptoms causing inability to perform usual social & functional activities OR Uncontrolled despite treatment modification | Life-threatening consequences (eg, myxedema coma) |
| Lipoatrophy (eg, fat loss from the face, extremities, buttocks) | Detectable by study<br>participant or caregiver<br>(for young children and<br>disabled adults) | Detectable on physical exam by health care provider | Disfiguring OR Obvious on casual visual inspection | NA |

| GENITOURINARY | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Intermenstrual Bleeding (IMB) | Spotting observed by participant<br>OR Minimal blood observed<br>during clinical or colposcopic<br>exam | Intermenstrual bleeding not greater in duration or amount than usual menstrual cycle | Intermenstrual bleeding greater in duration or amount than usual menstrual cycle | Hemorrhage with life-<br>threatening hypotension OR<br>Operative intervention<br>indicated |
| Urinary Tract<br>obstruction (eg, stone) | NA | Signs or symptoms of urinary tract obstruction without hydronephrosis or renal dysfunction | Signs or symptoms of urinary tract obstruction with hydronephrosis or renal dysfunction | Obstruction causing life-<br>threatening consequences |

| INFECTION | | | | |
|---|---|---|---|---|
| | Grade 1 | Grade 2 | Grade 3 | Grade 4 |
| Infection (any other than HIV infection) | Localized, no systemic antiµbial treatment indicated AND Symptoms causing no or minimal interference with usual social & functional activities | Systemic antiubial treatment indicated OR Symptoms causing greater than minimal interference with usual social & functional activities | Systemic antiubial treatment indicated AND Symptoms causing inability to perform usual social & functional activities OR Operative intervention (other than simple incision and drainage) indicated | Life-threatening consequences (eg, septic shock) |

Basic Self-care Functions: Activities such as bathing, dressing, toileting, transfer/movement, continence, and feeding.
Usual Social & Functional Activities: Adaptive tasks and desirable activities, such as going to work, shopping, cooking, use of transportation, pursuing a hobby, etc.

# Appendix 4. Pregnancy Precautions, Definition for Female of Childbearing Potential, and Contraceptive Requirements

### 1) Background

#### a) Ribavirin Warnings for Pregnancy

Ribavirin is contraindicated in pregnancy as significant teratogenic and embryocidal effects have been demonstrated in all animal species tested. Pregnancy must be excluded before the start of treatment with study drugs and prevented thereafter by reliable contraceptive methods. Pregnancy tests will be performed regularly throughout this study. Furthermore, RBV is known to accumulate intracellularly where it is cleared slowly, and is also excreted in semen. Therefore, extreme care must be taken to avoid pregnancy during RBV therapy and for 6 months following completion of treatment. Please refer to the latest version of the REBETOL® product insert for additional information

#### 2) Definitions

#### a) Definition of Childbearing Potential

For the purposes of this study, a female born subject is considered of childbearing potential following menarche until becoming post-menopausal, unless permanently sterile or with medically documented ovarian failure.

Women are considered to be in a postmenopausal state when they are  $\geq 54$  years of age with cessation of previously occurring menses for  $\geq 12$  months without an alternative cause.

Permanent sterilization includes hysterectomy, bilateral oophorectomy, or bilateral salpingectomy in a female subject of any age.

#### b) Definition of Male Fertility

For the purposes of this study, a male born subject is considered of fertile after the initiation of puberty unless permanently sterile by bilateral orchidectomy or medical documentation.

## 3) Study Drug Effect on Pregnancy and Hormonal Contraception

Data from clinical pharmacokinetic interaction studies of SOF have demonstrated that there is no reduction in the clinical efficacy of hormonal contraception. Non-clinical toxicity studies of SOF have demonstrated no adverse effect on fertility or embryo-fetal development.

Data from clinical pharmacokinetic interaction studies of VEL have demonstrated that there is no reduction in the clinical efficacy of hormonal contraception. Non-clinical toxicity studies of VEL have demonstrated no adverse effect on fertility or embryo-fetal development.

However, the risks of treatment with SOF/VEL during pregnancy in humans have not been evaluated. Please refer to the latest version of the Investigator's Brochure for additional information.

#### 4) Contraception Requirements for Female Subjects of Childbearing Potential

The inclusion of female subjects of childbearing potential requires using at least an acceptable effective contraceptive measure. They must have a negative serum pregnancy test at Screening and a negative pregnancy test on the Day 1 visit prior to first dose of study drug. Pregnancy testing will occur at regular intervals throughout the duration of the trial. In the event of a delayed menstrual period (over one month between menstruations), a pregnancy test must be performed to rule out pregnancy. This is even true for women of childbearing potential with infrequent or irregular periods. They must also agree to one of the following from Screening until 30 days after the last dose of SOF/VEL or 6 months after the last dose of RBV, whichever occurs last

• Complete abstinence from intercourse of reproductive potential. Abstinence is an acceptable method of contraception only when it is in line with the subject's preferred and usual lifestyle.

#### Or

- Consistent and correct use of 1 of the following methods of birth control listed below, in addition to a male partner who correctly used a condom from the date of Screening until 30 days after the last dose of SOF/VEL or 6 months after the last dose of RBV, whichever occurs last.
  - Intrauterine device (IUD)
  - Intrauterine hormone-releasing system (IUS)
  - Tubal sterilization
  - Essure micro-insert system (unapproved in Japan)
  - Vasectomy in the male partner
  - Barrier methods
    - Female barriers: Diaphragm with spermicide or Cervical cap with spermicide (unapproved in Japan)
  - Hormonal methods
    - Oral contraceptives (either combined or progesterone only)
    - Injectable progesterone (unapproved in Japan)
    - Implants of levonorgestrel or etonorgestrel (unapproved in Japan)
    - Transdermal contraceptive patch (unapproved in Japan)

#### ■ Contraceptive vaginal ring (unapproved in Japan)

Female subjects must also refrain from egg donation and in vitro fertilization during study treatment and until at least 30 days after the last dose of SOF/VEL or 6 months after the last dose of RBV, whichever occurs last.

#### 5) Contraception Requirements for Male Subjects

During the study, male subjects with female partners of childbearing potential should use condoms until 30 days after the last dose of SOF/VEL treatment or 6 months after the last dose of RBV, whichever comes last, when engaging in intercourse of reproductive potential. If their female partner is of childbearing potential (as defined above), their female partner must use 1 of the methods of birth control listed above from the date of Screening until 30 days after the last dose of SOF/VEL or 6 months after last dose of RBV, whichever comes last.

Male subjects must also refrain from sperm donation during treatment and until at least 30 days after the last dose of SOF/VEL or 6 months after the last dose of RBV, whichever comes last.

#### 6) Unacceptable Birth Control Methods

Birth control methods that are unacceptable include periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods), withdrawal (coitus interruptus), spermicides only, and lactational amenorrhea method (LAM). Female condom and male condom should not be used together.

#### 7) Procedures to be Followed in the Event of Pregnancy

Subjects will be instructed to notify the investigator if they become pregnant at any time during the study, if they become pregnant within 30 days of last dose of SOF/VEL, or if they become pregnant within 6 months of the last dose of RBV. Subjects who become pregnant or who suspect that they are pregnant during the study must report the information to the investigator and discontinue study drug immediately. Subjects whose partner has become pregnant or suspects she is pregnant within 30 days of the last dose of SOF/VEL or 6 months after the last dose of RBV, whichever occurs last, must report the information to the investigator.

Instructions for reporting pregnancy, partner pregnancy, and pregnancy outcome are outlined in Section 7.6.2.1.